CLINICAL TRIAL: NCT01975376
Title: Phase 3 Multi-center, Double-blind, Randomized, Placebo-controlled, Parallel Group Evaluation Of The Efficacy, Safety, And Tolerability Of Bococizumab (Pf-04950615) In Reducing The Occurrence Of Major Cardiovascular Events In High Risk Subjects.
Brief Title: The Evaluation of Bococizumab (PF-04950615;RN316) in Reducing the Occurrence of Major Cardiovascular Events in High Risk Subjects
Acronym: SPIRE-1
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: See Detailed Description
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B1481022; CV OUTCOMES 1; 2013-002646-36 (EudraCT Number); CV OUTCOMES 2 (Other: Alias Study Number)
Record Dates: First submitted 2013-10-21; First posted 2013-11-04 (Estimated); Results first posted 2018-06-12 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-06

CONDITIONS: Cardiovascular Disease
Keywords: myocardial infarction; stroke; hyperlipidemia
MeSH Terms: conditions — Cardiovascular Diseases; Myocardial Infarction; Stroke; Hyperlipidemias | interventions — bococizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- bococizumab (PF-04950615) (Experimental): 150 mg, every 2 weeks, subcutaneous
  Interventions: Drug: bococizumab (PF-04950615)
- Placebo (Placebo Comparator): Placebo comparator, every 2 weeks, subcutaneous.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: bococizumab (PF-04950615) — 150 mg, every 2 weeks, subcutaneous. The duration of the treatment period will depend upon reaching the targeted number of adjudicated and confirmed CV outcome events, approximately 3 to 4 years after the entry of first subject into the study.
  Other Names: RN316
  Arms: bococizumab (PF-04950615)
Drug: Placebo — Placebo comparator, every 2 weeks, subcutaneous. The duration of the treatment period will depend upon reaching the targeted number of adjudicated and confirmed CV outcome events, approximately 3 to 4 years after the entry of first subject into the study.
  Arms: Placebo

SUMMARY:
This study evaluates the PCSK9 inhibitor, Bococizumab (PF-04950615;RN316), compared to placebo, in reducing the occurrence of major cardiovascular events, including cardiovascular death, myocardial infarction, stroke, and unstable angina requiring urgent revascularization, in high risk subjects who are receiving background lipid lowering therapy and have cholesterol laboratory values of LDL-C >/= 70 mg/dL (1.8 mmol/L) or non-HDL-C >/= 100 mg /dL (2.6 mmol/L).

DETAILED DESCRIPTION:
The trial was terminated prematurely on November 1, 2016, due to the emerging clinical profile and the evolving treatment and market landscape for lipid-lowering agents. These indicated that bococizumab was not likely to provide value to patients, physicians, or shareholders. The decision was not based on a recommendation by the independent Data Monitoring Committee to stop the program.

ELIGIBILITY:
Inclusion Criteria:

* Must be on background lipid lowering treatment.
* Must be at high risk of a CV event.
* Must have an LDL C >/=70 mg/dL (1.8 mmol/L) or non-HDL-C >/= 100 mg/dL (2.6 mmol/L).

Exclusion Criteria:

* Planned coronary (PCI or CABG) or other arterial revascularization.
* New York Heart Association Class IV congestive heart failure or left ventricular ejection fraction < 25% by cardiac imaging.
* Chronic renal insufficiency with creatinine clearance of <30 ml/min/1.73m^2 by MDRD formula or with end state renal disease on dialysis.
* History of hemorrhagic stroke.
* Prior exposure to bococizumab or other investigational PCSK9 inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16784 (Actual)
Dates: Start 2013-10-29 (Actual); Primary Completion 2017-03-22 (Actual); Study Completion 2017-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1740):
- United States (543):
  - Ernest Hendrix, MD, PC, Athens, Alabama
  - North Alabama Research Center LLC, Athens, Alabama
  - Central Alabama Research, Birmingham, Alabama
  - Clinical Research Advantage, Inc./Simon Williamson Clinic, Birmingham, Alabama
  - Birmingham Heart Clinic, P.C., Birmingham, Alabama
  - Cardiovascular Associates of the Southeast, LLC, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Appalachian Cardiovascular Associates, Fort Payne, Alabama
  - Fundamental Research, LLC, Gulf Shores, Alabama
  - Avant Research Associates, LLC, Guntersville, Alabama
  - Boyett Health Services, Hamilton, Alabama
  - Saadat Ansari Internal Medicine, Huntsville, Alabama
  - CB Flock Research Corporation, Mobile, Alabama
  - Alaska Heart Institute, Anchorage, Alaska
  - Phoenix Heart, PLLC, Glendale, Arizona
  - Arrowhead Internal Medicine, Glendale, Arizona
  - Clinical Research Advantage, Inc./Family Practice Specialists, Ltd., Phoenix, Arizona
  - Redpoint Research, Phoenix, Arizona
  - Cochise Clinical Research, Sierra Vista, Arizona
  - Clinical Research Advantage, Inc. (Administrative Mailing Only), Tempe, Arizona
  - Southwest Heart Group, Tucson, Arizona
  - University of Arizona Medical Center South Campus, Tucson, Arizona
  - Arizona Endocrine and Rheumatology Associates, Tucson, Arizona
  - Arkansas Heart Hospital Clinic, Little Rock, Arkansas
  - Arkansas Site Management Services, LLC, Little Rock, Arkansas
  - Cardiology Consultants of Orange County Medical Group Inc., Anaheim, California
  - Premier Valley Medical Group, Bakersfield, California
  - Cardiovascular Research Foundation of Southern California, Beverly Hills, California
  - Westside Medical Associates of Los Angeles, Beverly Hills, California
  - Southbay Pharma Research, Buena Park, California
  - Med Center, Carmichael, California
  - Pioneer Medical Group, Cerritos, California
  - John Muir Physician Network Clinical Research Center, Concord, California
  - Atlantic Ave Medical Clinic Inc., Cudahy, California
  - Multani Medical Group, Downey, California
  - Triwest Research Associates, LLC, El Cajon, California
  - Diagnamics, Inc., Encinitas, California
  - T. Joseph Raoof, Md, Inc/Encino Research Center, Encino, California
  - Aviva Research, Escondido, California
  - Med Investigations, Inc., Fair Oaks, California
  - Valley Research, Fresno, California
  - St. Jude Hospital Yorba Linda DBA St. Joseph Heritage Healthcare, Fullerton, California
  - Omnibus Clinical Research, La Palma, California
  - Alliance Research Centers, Laguna Hills, California
  - Prime Care Clinical Research Center, Laguna Hills, California
  - Clinical Trials Research, Lincoln, California
  - Long Beach Memorial Medical Center, Long Beach, California
  - American Institute of Research, Los Angeles, California
  - Intermed Group, Los Angeles, California
  - Academic Medical Research Institute, Los Angeles, California
  - Eastside Clinical Research Associates, Los Angeles, California
  - Richard S. Cherlin, MD, Los Gatos, California
  - Facey Medical Foundation, Mission Hills, California
  - California Medical Research Associates Inc., Northridge, California
  - Valley Clinical Trials, Inc., Northridge, California
  - Diabetes Associates Medical Group, Orange, California
  - Saviers Medical Group, Port Hueneme, California
  - Arch Health Partners, Poway, California
  - A. R. I. Clinical Trials, Inc., Redondo Beach, California
  - California Research Foundation, San Diego, California
  - San Diego Family Care dba Linda Vista Health Center, San Diego, California
  - San Diego Family Care, San Diego, California
  - Ritchken & First Md's, San Diego, California
  - Wetlin Research Associates, Inc., San Diego, California
  - West Coast Research LLC, San Ramon, California
  - Syrentis Clinical Research, Santa Ana, California
  - Coastal Biomedical Research, Inc., Santa Monica, California
  - Encompass Clinical Research, Spring Valley, California
  - St. Joseph's Medical Associates, Stockton, California
  - Westlake Medical Research, Thousand Oaks, California
  - Los Angeles Biomedical Research Institute at Harbor - UCLA Medical Center, Torrance, California
  - Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Torrance, California
  - Harbor - UCLA Medical Center, Torrance, California
  - Orange County Research Center, Tustin, California
  - Bayview Research Group, Valley Village, California
  - Coastal Metabolic Research Centre, Ventura, California
  - Ventura Clinical Trials, Ventura, California
  - Clinical Research Advantage, Inc. / Cassidy Medical Group - Vista, Vista, California
  - Allianz Research Institute, Westminster, California
  - American Institute of Research Studies, Whittier, California
  - Elite Clinical Trials, Inc., Wildomar, California
  - Elite Clinical Trials, Incorporated, Wildomar, California
  - Colorado Springs Health Partners, Colorado Springs, Colorado
  - ExpressCare Clinical Research, Colorado Springs, Colorado
  - Lynn Institute of the Rockies, Colorado Springs, Colorado
  - Memorial Hospital: University of Colorado Health, Colorado Springs, Colorado
  - Lynn Institute of Denver, Denver, Colorado
  - Western Colorado Research, LLC, Glenwood Springs, Colorado
  - South Denver Cardiology Associates, PC, Littleton, Colorado
  - Connecticut Clinical Research, LLC, Bridgeport, Connecticut
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Cardiology Associates of Fairfield County, PC, Stamford, Connecticut
  - Stamford Therapeutics Consortium, Stamford, Connecticut
  - Christiana Care Health Services, Inc., Newark, Delaware
  - Alfieri Cardiology, Wilmington, Delaware
  - Capital Medical Associates, PC, Washington D.C., District of Columbia
  - ACRC - Cardiology, Atlantis, Florida
  - Meridien Research, Brooksville, Florida
  - Gulf Coast Endocrine and Diabetes Center, Clearwater, Florida
  - Team Medical Research, Coral Gables, Florida
  - The Heart Group, PA, Daytona Beach, Florida
  - Cardiology Associates Research Company, Daytona Beach, Florida
  - Seidman Clinical Trials, Delray Beach, Florida
  - The Cardiology Center, Delray Beach, Florida
  - Continental Research Corp, Doral, Florida
  - Care Research Center Inc, Doral, Florida
  - Integrity Clinical Research, LLC, Doral, Florida
  - Moonshine Research Center, Inc., Doral, Florida
  - Advanced Clinical Research of Miami (ACROM) International, Doral, Florida
  - Invesclinic, LLC, Fort Lauderdale, Florida
  - The Office of Alan Graff, MD, PA, Fort Lauderdale, Florida
  - The Center for Diabetes and Endocrine Care, Fort Lauderdale, Florida
  - Broward Health Medical Center (BHMC) (Broward General Medical Center (BGMC)), Fort Lauderdale, Florida
  - The Office of Maxine E. Hamilton, MD, PA, Fort Lauderdale, Florida
  - State Of The Art Research, LLC, Hialeah, Florida
  - Direct Helpers Medical Center Inc, Hialeah, Florida
  - Research Physicians Network Alliance, Hollywood, Florida
  - Pines Clinical Research, Inc., Hollywood, Florida
  - East Coast Institute for Research, LLC, Jacksonville, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - River City Clinical Research, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Baker-Gilmore Cardiovascular Institute, Jacksonville, Florida
  - Solutions Through Advanced Research, Inc., Jacksonville, Florida
  - Meridien Research, Lakeland, Florida
  - The Heart Institute at Largo, Largo, Florida
  - South Florida Clinical Research Institute, Margate, Florida
  - Accelovance, Melbourne, Florida
  - Future Clinical Research, Inc., Miami, Florida
  - Advanced Clinical Research of Miami (ACROM) International, Miami, Florida
  - Project4Research, Inc, Miami, Florida
  - A & L Clinical Research, Miami, Florida
  - Finlay Medical Research, Miami, Florida
  - Pharmax Research Clinic, Inc., Miami, Florida
  - South Florida Research Center, Inc., Miami, Florida
  - Florida Medical Center & Research, Inc., Miami, Florida
  - Medical Research Center, Miami, Florida
  - Nuren Medical & Research Center, Miami, Florida
  - Doctors Research Institute, Miami, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - Coast Research Institute, Miami, Florida
  - My Community Research Center, Inc., Miami, Florida
  - Columbus Clinical Services LLC, Miami, Florida
  - Cardiovascular Research Center of South Florida, Miami, Florida
  - Research Institute of South Florida, Inc., Miami, Florida
  - A & O Research Center, Inc., Miami, Florida
  - BWell Research Center, Miami, Florida
  - Pharmacology International Research, Inc., Miami, Florida
  - Advanced Clinical Research, Miami, Florida
  - South Florida Research Group, LLC, Miami, Florida
  - International Research Associates, LLC, Miami, Florida
  - Kendall South Medical Center, Inc., Miami, Florida
  - M & M Medical Center, Inc, Miami, Florida
  - Med Research Of Florida, LLC, Miami, Florida
  - Research Physicians Network Alliance, Miami Beach, Florida
  - G & I Medical Research LLC, Miami Lakes, Florida
  - Southwest Florida Research, Naples, Florida
  - BayCare Medical Group, New Port Richey, Florida
  - The Heart & Vascular Institute of Florida, New Port Richey, Florida
  - Bravo Health Care Center, North Bay Village, Florida
  - Harmony Clincal Research, Inc., North Miami Beach, Florida
  - Florida Hospital Cardiovascular Institute, Orlando, Florida
  - Omega Research Consultants, LLC, Orlando, Florida
  - Aba Family Medicine, LLC, Ormond Beach, Florida
  - Millennium Research, Ormond Beach, Florida
  - Ribo Research, LLC dba Peninsula Research, Ormond Beach, Florida
  - A&R Research Group, LLC, Pembroke Pines, Florida
  - Research Physicians Network Alliance, Pembroke Pines, Florida
  - South Broward Research, Pembroke Pines, Florida
  - DBC Research USA, Pembroke Pines, Florida
  - DBC Research, Pembroke Pines, Florida
  - Cardiology Consultants, Pensacola, Florida
  - DMI Research, Inc., Pinellas Park, Florida
  - Clincal Research of Florida, Plant City, Florida
  - Clinical Research of Central Florida, Plant City, Florida
  - Dr. Jeffrey Greiff MD, Office Of, Plantation, Florida
  - Nova Clinical Research Collaborative, Plantation, Florida
  - St. Johns Center for Clinical Research, Ponte Vedra, Florida
  - Charlotte Heart Group Research Center, Port Charlotte, Florida
  - Intercoastal Medical Group, Sarasota, Florida
  - Cardiovascular Center Of Sarasota, Sarasota, Florida
  - Heart & Vascular Center Research, Sarasota, Florida
  - Intercoastal Medical Group (Drug Shipment Address and Administrative), Sarasota, Florida
  - The Office of Bridget Bellingar, DO, Seminole, Florida
  - Meridien Research, St. Petersburg, Florida
  - Advance Medical Research, St. Petersburg, Florida
  - Vita Health & Medical Center, Inc./Concept Clinical Trials, LLC, Tamarac, Florida
  - Interventional Cardiac Consultants, Trinity, Florida
  - Cardiology Partners Clinical Research Institute, Wellington, Florida
  - Cleveland Clinic Cardiology Associates, West Palm Beach, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Clinical Research of Central Florida, Winter Haven, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Atlanta Center For Medical Research, Atlanta, Georgia
  - Columbus Regional Research Institute, Columbus, Georgia
  - Rockdale Medical Research Associates, Conyers, Georgia
  - Georgia Heart Specialists, LLC, Covington, Georgia
  - Neurostudies.Net, LLC, Decatur, Georgia
  - Alta Pharmaceutical Research Center, Dunwoody, Georgia
  - In-Quest Medical Research, LLC, Norcross, Georgia
  - Atlanta Center for Clinical Research / Internal Medicine, Roswell, Georgia
  - Dr. B. Abraham, P.C., Snellville, Georgia
  - Georgia Clinical Research, LLC, Snellville, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Elite Clinial Trials, LLLP, Blackfoot, Idaho
  - Elite Clinial Trials, Blackfoot, Idaho
  - St. Luke's Idaho Cardiology Associates, Caldwell, Idaho
  - Solaris Clinical Research, Meridian, Idaho
  - Saltzer Medical Group, PA, Nampa, Idaho
  - Northwest Heart Clinical Research, LLC, Arlington Heights, Illinois
  - Clinical Research Advantage, Inc./Michigan Avenue Internists, Chicago, Illinois
  - Apex Medical Research, AMR, Inc., Chicago, Illinois
  - Clinical Research Advantage, Inc./Medical and Procedural Specialists of Illinois, Chicago, Illinois
  - Evanston Premier Healthcare Research, LLC, Evanston, Illinois
  - Clinical Investigation Specialists, Inc, Gurnee, Illinois
  - Heart Care Centers of Illinois, Mokena, Illinois
  - Advanced CardioVascular Consultants, Rock Island, Illinois
  - Investigators Research Group, LLC, Brownsburg, Indiana
  - Investigative Clinical Research of Indiana, LLC, Elwood, Indiana
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Clinical Research Advantage, Inc. (IP Shipment and Research Site), Evansville, Indiana
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Clinical Research Advantage, Inc. / Family Medicine Associates, Evansville, Indiana
  - Deaconess Clinic Mt. Pleasant, Evansville, Indiana
  - American Health Network of Indiana LLC, Franklin, Indiana
  - American Health Network of Indiana, LLC, Greenfield, Indiana
  - American Health Network of Indiana, LLC, Muncie, Indiana
  - Cardiovascular Research of Northwest Indiana, LLC, Munster, Indiana
  - Buynak Clinical Research, P.C., Valparaiso, Indiana
  - West Broadway Clinic, Council Bluffs, Iowa
  - Clinical Research Advantage, Inc., Council Bluffs, Iowa
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - University of Iowa College of Public Health - Preventive Intervention Center, Iowa City, Iowa
  - Northeast Iowa Medical Education Foundation, Waterloo, Iowa
  - The Iowa Clinic, PC, West Des Moines, Iowa
  - Hutchinson Clinic, P.A, Hutchinson, Kansas
  - University Of Kansas Medical Center, Kansas City, Kansas
  - Heartland Research Associates, LLC, Newton, Kansas
  - Midwest Heart & Vascular Specialists, LLC, Overland Park, Kansas
  - Women's & Family Care, LLC D.B.A GTC Research, Shawnee Mission, Kansas
  - Central Cardiology Associates Research, Elizabethtown, Kentucky
  - The Research Group of Lexington, LLC, Lexington, Kentucky
  - L-MARC Research Center, Louisville, Kentucky
  - Research Integrity, LLC., Owensboro, Kentucky
  - Alexandria Cardiology Clinic, Alexandria, Louisiana
  - Avant Research Associates, LLC, Crowley, Louisiana
  - Centex Studies, Lake Charles, Louisiana
  - Imperial Health, LLC, Lake Charles, Louisiana
  - American Clinical Research, LLC, Marrero, Louisiana
  - West Jefferson Heart Clinic of Louisiana New Orleans Physician Services, Inc., Marrero, Louisiana
  - Clinical Trials of America LA, Monroe, Louisiana
  - KAMP Medical Research Inc., Natchitoches, Louisiana
  - Grace Research, LLC, Shreveport, Louisiana
  - Maine Research Associates, Auburn, Maine
  - Acadia Clinical Research, LLC, Bangor, Maine
  - Cranbrook Cardiology Research Associates, Westbrook, Maine
  - Anne Arundel Medical Center, Annapolis, Maryland
  - MedStar Cardiology Associates, Annapolis, Maryland
  - MedStar Chesapeake CardioVascular Associates, Baltimore, Maryland
  - MedStar Union Memorial Heart Specialists, Baltimore, Maryland
  - Maryland Cardiovascular Specialists, Baltimore, Maryland
  - Overlea Personal Physicians, Baltimore, Maryland
  - Shahid Saeed, MD, PC, Baltimore, Maryland
  - Maryland Heart Associates, LLC, Glen Burnie, Maryland
  - Lutherville Personal Physicians, Lutherville, Maryland
  - MD Medical Research, Oxon Hill, Maryland
  - Metro West Medical Center Research Clinic, Framingham, Massachusetts
  - Metro West Medical Center, Framingham, Massachusetts
  - MetroWest Medical Center - Pharmacy Department, Framingham, Massachusetts
  - Pentucket Medical Associates, LLC, Haverhill, Massachusetts
  - ActivMed Practices and Research, Inc., Methuen, Massachusetts
  - Charles River Medical Associates, Natick, Massachusetts
  - Endeavor Medical Research, Alpena, Michigan
  - St. Joseph Mercy Health System, Ann Arbor, Michigan
  - University of Michigan - Domino Farms, Ann Arbor, Michigan
  - IHA Chelsea Family & Internal Medicine, Chelsea, Michigan
  - Healthy Heart Cardiology, Grandville, Michigan
  - Westside Family Medical Center, Pc, Kalamazoo, Michigan
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Sparrow Thoracic & Cardiovascular Institute, Lansing, Michigan
  - Detroit Clinical Research Center, PC, Livonia, Michigan
  - MidMichigan Medical Center Midland, Midland, Michigan
  - Michigan Cardio Vascular Institute, Saginaw, Michigan
  - Tri-County Research, Inc., Sterling Heights, Michigan
  - Medical Research Associates, Inc., Traverse City, Michigan
  - Oakland Medical Research Center, Troy, Michigan
  - Arcturus Healthcare, PLC, Troy Internal Medicine Research Division, Troy, Michigan
  - Michigan Heart & Vascular Institute, Ypsilanti, Michigan
  - Duluth Clinic, dba Essentia Health Duluth Clinic Investigational Drug Room, Duluth, Minnesota
  - St. Mary's Medical Center (Primary Practice Site), Duluth, Minnesota
  - Radiant Research, Inc., Edina, Minnesota
  - Minneapolis Clinic of Neurology, Golden Valley, Minnesota
  - Allina Health System, dba Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Lillehei Clinical Research Unit, University of Minnesota, Minneapolis, Minnesota
  - CentraCare Heart and Vascular Center, Saint Cloud, Minnesota
  - HealthEast Medical Research Institute, Saint Paul, Minnesota
  - HealthEast St. Joseph's Hospital Pharmacy, Saint Paul, Minnesota
  - Phillips Medical Services, PLLC, Jackson, Mississippi
  - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - Cardiology Associates Research, LLC, Tupelo, Mississippi
  - Missouri Cardiovascular Specialists, LLP, Columbia, Missouri
  - Saint Luke's Lipid and Diabetes Research Center, Kansas City, Missouri
  - Kansas City VA Medical Center, Kansas City, Missouri
  - Mercy Research, St Louis, Missouri
  - Glacier View Research Institute, Kalispell, Montana
  - Glacier View Research Institute, Cardiology, Kalispell, Montana
  - Montana Medical Research Inc., Missoula, Montana
  - Clinical Research Advantage, Inc./Skyline Medical Center, PC, Elkhorn, Nebraska
  - Bryan Heart, Lincoln, Nebraska
  - Creighton Diabetes Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - AB Clinical Trials, Las Vegas, Nevada
  - Clinical Research Of South Nevada, Las Vegas, Nevada
  - Clinical Research Advantage, Inc., Las Vegas, Nevada
  - John V. Bernard, MD dba Wellness and Research Center, Belvidere, New Jersey
  - Advanced Heart Care LLC, Bridgewater, New Jersey
  - Lourdes Cardiology Services, Cherry Hill, New Jersey
  - USMA Clinical Research, Elizabeth, New Jersey
  - Lourdes Cardiology Services, Hammonton, New Jersey
  - NJ Heart, Linden, New Jersey
  - Arysmed LLC, Lodi, New Jersey
  - Amici Clinical Research, LLC, Martinsville, New Jersey
  - Rutgers Biomedical and Health Sciences-Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Cardiac and Endovascular Associates, Ridgewood, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Cardio Metabolic Institute, Somerset, New Jersey
  - TLB Research LLC, Trenton, New Jersey
  - Lourdes Cardiology Services, Voorhees Township, New Jersey
  - Westwood Cardiology Associates, Westwood, New Jersey
  - Albuquerque Clinical Trials, Inc., Albuquerque, New Mexico
  - Albany Medical College, Division of Community Endocrinology, Albany, New York
  - Sorin Medical, P.C., Brooklyn, New York
  - NY Total Medical Care, PC, Brooklyn, New York
  - NY Scientific, Brooklyn, New York
  - Buffalo Heart Group, Llp, Buffalo, New York
  - NYU Hudson Valley Cardiology, Cortlandt Manor, New York
  - Scott Research,Inc, Laurelton, New York
  - SJH Cardiology Associates, Liverpool, New York
  - Long Island Heart Associates, Mineola, New York
  - Mid Hudson Medical Research, PLLC, New Windsor, New York
  - Manhattan Medical Research Practice, New York, New York
  - Peters Medical Research NY, LLC, New York, New York
  - Weill Cornell Medical College, New York, New York
  - DiGiovanna Institute for Medical Education And Research, North Massapequa, New York
  - Hudson Valley Cardiovascular Practice, PC, Poughkeepsie, New York
  - Rochester Clinical Research, Inc., Rochester, New York
  - Institute for Clinical Studies, Rosedale, New York
  - Saratoga Clinical Research, LLC, Saratoga Springs, New York
  - Central New York Cardiology, Utica, New York
  - Great Lakes Medical Research, Westfield, New York
  - Buffalo Medical Group - Research Department, Williamsville, New York
  - Buffalo Medical Group, Williamsville, New York
  - Kernodle Clinic, Department of the Private Diagnostic Clinic, PLLC, Burlington, North Carolina
  - Novant Health Clinical Research, Charlotte, North Carolina
  - Novant Health Heart and Vascular Institute, Charlotte, North Carolina
  - PMG Research of Charlotte, Charlotte, North Carolina
  - Sensenbrenner Primary Care, Charlotte, North Carolina
  - NC Heart and Vascular, Clayton, North Carolina
  - LeBauer Cardiovascular Research Foundation, Greensboro, North Carolina
  - Clinical Trials of America, Inc., Hickory, North Carolina
  - Carolina Cardiology Cornerstone, High Point, North Carolina
  - Clinical Trials of America- NC, LLC, Lenoir, North Carolina
  - Research Institute of the Carolinas of PiedmontHealthcare, PA, Mooresville, North Carolina
  - Burke Primary Care, Morganton, North Carolina
  - Eastern Nephrology Associates, New Bern, North Carolina
  - Boice Willis Clinic, Rocky Mount, North Carolina
  - PMG Research of Rock Mount, LLC - Patient Intake, Rocky Mount, North Carolina
  - Piedmont Healthcare/Research, Statesville, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Radiant Research, Inc., Akron, Ohio
  - The Lindner Center for Research and Education at The Christ Hospital, Cincinnati, Ohio
  - Metabolic and Atherosclerosis Research Center, Cincinnati, Ohio
  - Sterling Research Group, Ltd., Cincinnati, Ohio
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Cleveland Clinic - Taussig Cancer Institute, Cleveland, Ohio
  - Radiant Research, Inc., Columbus, Ohio
  - Optimed Research, LTD, Columbus, Ohio
  - Premier Health Specialists, Inc (dba Dayton Heart Center), Dayton, Ohio
  - PriMed Clinical Research, Dayton, Ohio
  - North Ohio Heart Center (Administrative Only), Elyria, Ohio
  - North Ohio Heart Center, Elyria, Ohio
  - North Ohio Heart Center, Lorain, Ohio
  - SV Research, LLC, Marion, Ohio
  - Daniel G. Williams, MD, Perrysburg, Ohio
  - North Ohio Heart Center, Inc., Sandusky, Ohio
  - North Ohio Heart Center, Sandusky, Ohio
  - ProMedica Northwest Ohio Cardiology Consultants, Toledo, Ohio
  - Mercy Health Youngstown, LLC d/b/a St. Elizabeth Youngstown Hospital, Youngstown, Ohio
  - LION Research, Norman, Oklahoma
  - COR Clinical Research LLC, Oklahoma City, Oklahoma
  - Oklahoma Heart Hospital Physicians, Oklahoma City, Oklahoma
  - Oklahoma Heart Hospital Research Foundation, Oklahoma City, Oklahoma
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - South Oklahoma Heart Research, LLC, Oklahoma City, Oklahoma
  - Integrated Medical Research PC, Ashland, Oregon
  - Hillsboro Cardiology, P.C., Hillsboro, Oregon
  - Portland Preventive Cardiology LLC, Portland, Oregon
  - Abington Memorial Hospital (administrative only), Abington, Pennsylvania
  - Clinical Research Associates of Central PA, Altoona, Pennsylvania
  - Brandywine Clinical Research, Downingtown, Pennsylvania
  - Doylestown Cardiology Associates - VIAA, Doylestown, Pennsylvania
  - Doylestown Health Cardiology, a division of Doylestown Health Physicians, Doylestown, Pennsylvania
  - AMH/Feasterville Family Health Care Center, Feasterville-Trevose, Pennsylvania
  - Greater Pittsburgh Vascular, Jefferson Hills, Pennsylvania
  - Detweiler Family Medicine & Associates, PC, Lansdale, Pennsylvania
  - Green and Seidner Family Practice Associates, Lansdale, Pennsylvania
  - Family Medical Associates, Levittown, Pennsylvania
  - Mercer Bucks Cardiology, Newtown, Pennsylvania
  - Philadelphia Health Associates-Adult Medicine, Philadelphia, Pennsylvania
  - Allegheny Endocrinology Associates, Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Pittsburgh, Pennsylvania
  - Guthrie Medical Group, PC, Sayre, Pennsylvania
  - SFM Clinical Trials, Inc., Scotland, Pennsylvania
  - Fay-West Family Practice, Scottdale, Pennsylvania
  - Grand View - Lehigh Valley Health Services, Buxmont Cardiology Division, Sellersville, Pennsylvania
  - Montgomery Medical, Inc., Smithfield, Pennsylvania
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - Berks Cardiologists, Ltd., Wyomissing, Pennsylvania
  - Coastal Cardiolgy, Charleston, South Carolina
  - Upstate Pharmaceutical Research, Greenville, South Carolina
  - Mountain View Clinical Research, Inc., Greer, South Carolina
  - Black Hills Cardiovascular-Regional Health Research, Rapid City, South Dakota
  - Mid-Cumberland Infectious Disease Consultants, PLC, Clarksville, Tennessee
  - Collierville Medical Specialists, Collierville, Tennessee
  - Stern Cardiovascular Foundation, Inc., Germantown, Tennessee
  - Holston Medical Group, Kingsport, Tennessee
  - New Phase Research & Development, Knoxville, Tennessee
  - PMG Research,Inc d/b/a PMG Research of Knoxville, Knoxville, Tennessee
  - Cardiovascular Research of Knoxville, Knoxville, Tennessee
  - New Orleans Center for Clinical Research, Knoxville, Tennessee
  - Volunteer Research Group, Knoxville, Tennessee
  - Baptist Memorial Medical Group, Inc., Memphis, Tennessee
  - The Green Clinic, PC, Memphis, Tennessee
  - Southwind Medical Specialists, Memphis, Tennessee
  - Tennessee Center for Clinical Trials, Tullahoma, Tennessee
  - Trinity Clinical Research, LLC, Tullahoma, Tennessee
  - PharmaTex Research, Amarillo, Texas
  - Arlington Family Research Center, Inc., Arlington, Texas
  - Texas Diabetes & Endocrinology, Austin, Texas
  - Austin Heart, PLLC, Austin, Texas
  - Southeast Texas Cardiology Associates II, L.L.P., Beaumont, Texas
  - Southeast Texas Clinical Research Center, Beaumont, Texas
  - Aztec Medical Research, LLC, Channelview, Texas
  - Corsicana Medical Research, PLLC, Corsicana, Texas
  - Baylor Research Institute IRB, Dallas, Texas
  - Protenium Clinical Research, LLC, Dallas, Texas
  - VA North Texas Health Care System - Dallas VAMC, Dallas, Texas
  - Baylor Heart and Vascular Institute, Dallas, Texas
  - Dallas Diabetes and Endocrine Center, Dallas, Texas
  - Cardiovascular Research Institute of Dallas, Dallas, Texas
  - Radiant Research, Inc., Dallas, Texas
  - Research Institute of Dallas, Dallas, Texas
  - Parkland Health and Hospital System, Dallas, Texas
  - Baylor University Medical Center / Department of Pharmacy, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - (For IP storage only)The University of Texas Southwestern Medical Center, Dallas, Texas
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - William P. Clements Jr. University Hospital, Dallas, Texas
  - Doctors Hospital At Renaissance, Edinburg, Texas
  - Amir Malik Research, Fort Worth, Texas
  - The Medical Group of Texas, Fort Worth, Texas
  - T & R Clinic, PA, Fort Worth, Texas
  - Rockwood Medical Clinic, Fort Worth, Texas
  - San Gabriel Clinical Research, LLC, Georgetown, Texas
  - East Texas Cardiology PA, Houston, Texas
  - Spring Clinical Research, Houston, Texas
  - Med Tech Research, LP, Houston, Texas
  - Prime Care Medical Group, Houston, Texas
  - Associates in Medicine, PA, Houston, Texas
  - Alan S. Hoffman, M.D., Houston, Texas
  - Baylor College of Medicine, Houston, Texas
  - ICTR/Baylor College of Medicine, Houston, Texas
  - Investigational Drug Services, Houston, Texas
  - Memorial Hermann Hospital, Texas Medical Center- UT Health Clinical Research Unit, Houston, Texas
  - Memorial Hermann Hospital, Texas Medical Center, Houston, Texas
  - The University of Texas Health Science Center at Houston- UT Physicians, Houston, Texas
  - Centex Studies, Inc., Houston, Texas
  - Northwest Houston Cardiology, P.A., Houston, Texas
  - Texas Center for Drug Development, Inc, Houston, Texas
  - Private Practice Leadership, LLC, Houston, Texas
  - Protenium Clinical Research LLC, Hurst, Texas
  - South Texas Cardiovascular Consultants, PLLC, Kerrville, Texas
  - DCOL Center for Clinical Research, Longview, Texas
  - Caprock Cardiac Center Research Institute Inc., Lubbock, Texas
  - Midland Clinical Research Center, Midland, Texas
  - Hill Country Medical Associates, New Braunfels, Texas
  - North Hills Medical Research, Inc., North Richland Hills, Texas
  - Grace Research, LLC, Palestine, Texas
  - Med-Olam Clinical Research, LLC., Pasadena, Texas
  - Austin Institute for Clinicla Research,Inc., Pflugerville, Texas
  - Centex Studies, Inc, Pharr, Texas
  - South Texas Cardiovascular Consultants, PLLC, San Antonio, Texas
  - Sun Research Institute, San Antonio, Texas
  - Southwest Clinic, San Antonio, Texas
  - FIRST Outpatient Research Unit, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - University of Texas Health Science Center San Antonio, San Antonio, Texas
  - University of Texas Health Sciences Center at San Antonio, San Antonio, Texas
  - Victorium Clinical Research, San Antonio, Texas
  - Bandera Family Health Care, LLC, San Antonio, Texas
  - Northeast Clinical Research of San Antonio, LLC (NECRSA, LLC), Schertz, Texas
  - Acacia Medical Research Institute, LLC/Royal Oaks Medcical Home and Wellness Clinics, Sugar Land, Texas
  - IP + Dry ice deliveries Sugar Lakes Family Practice, Sugar Land, Texas
  - Sugar Lakes Family Practice, Sugar Land, Texas
  - Northwest Houston Heart Center, Tomball, Texas
  - Admin & Storage only:Northwest Heart Center, Tomball, Texas
  - Northwest Heart Center, Tomball, Texas
  - Northwest Houston Clinical Research, PLLC, Tomball, Texas
  - Victoria Heart & Vascular Center, PA, Victoria, Texas
  - Victoria Heart and Vascular Center, PA, Victoria, Texas
  - Utah Cardiology, PC, Bountiful, Utah
  - Utah Cardiology, P.C., Layton, Utah
  - Paramount Medical Care, Ogden, Utah
  - Aspen Clinical Research LLC, Orem, Utah
  - Revere Health, Provo, Utah
  - Optimum Clinical Research, Inc, Salt Lake City, Utah
  - Wasatch Clinical Research, LLC, Salt Lake City, Utah
  - Holladay Family Practice, Salt Lake City, Utah
  - Heart Center at St. Mark's Hospital, Salt Lake City, Utah
  - Clinical Research Institute of Northern Virginia, Burke, Virginia
  - Burke Internal Medicine & Research, Burke, Virginia
  - Virginia Heart, Falls Church, Virginia
  - Seven Corners Medical Research Center, Falls Church, Virginia
  - Heart Care Associates, P.C., Hopewell, Virginia
  - Virginia Research Center, Midlothian, Virginia
  - Chippenham and Johnston Willis Hospitals, Inc. dba CJW Medical Center, Richmond, Virginia
  - Retreat Cardiology LLC, dba Cardiology Associates of Richmond, Richmond, Virginia
  - Roanoke Heart Institute, Roanoke, Virginia
  - Hampton Roads Center for Clinical Research, Suffolk, Virginia
  - The Office of Daniel W. Gottlieb, MD, PS, Burien, Washington
  - Premier Clinical Research, Spokane, Washington
  - Universal Research Group, LLC, Tacoma, Washington
  - Walla Walla Clinic, Walla Walla, Washington
  - Wenatchee Valley Hospital & Clinics, Wenatchee, Washington
  - Fairmont General Hospital, Fairmont, West Virginia
  - Prevea Clinic, Inc., Green Bay, Wisconsin
  - Clinical Investigation Specialists, Inc., Kenosha, Wisconsin
  - Waukesha Heart Foundation, Waukesha, Wisconsin
- Argentina (48):
  - Instituto de Investigaciones Clinicas Bahia Blanca, Bahía Blanca, Buenos Aires
  - Hospital Italiano Regional del Sur, Bahía Blanca, Buenos Aires
  - Hospital Britanico De Buenos Aires, Ciudad Autonoma de B. Aires, Buenos Aires
  - CEDIC - Consultorios Medicos, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Clinica Coronel Suarez S.A., Coronel Suárez, Buenos Aires
  - Framingham Centro Medico, La Plata, Buenos Aires
  - CIMeL CHAHIN CHAHIN S.A., Lanús Este, Buenos Aires
  - Instituto de Investigaciones Clinicas Mar del Plata, Mar del Plata, Buenos Aires
  - Instituto de Investigaciones Clinicas Quilmes, Quilmes, Buenos Aires
  - DIM Clinica Privada, Ramos Mejía, Buenos Aires
  - Instituto de Investigaciones Clinicas Zarate, Zárate, Buenos Aires
  - STAT Research S.A., C.a.b.a, Buenos Aires F.D.
  - Consultorios Asociados de Endocrinologia e Investigacion Clinica Aplicada, C.a.b.a, C.a.b.a.
  - Clinica Privada de Especialidades Medicas, Villa María, Córdoba Province
  - CIPADI Centro Integral de Prevencion y Atencion en Diabetes, Godoy Cruz, Mendoza Province
  - Hospital Interzonal Gral. de Agudos Dr. Jose Penna, Bahía Blanca, PCIA de Buenos Aires
  - IMEP Instituto Medico Elsa Perez, Ciudadela, PCIA de Buenos Aires
  - Instituto Medico Aguero, Morón, PCIA de Buenos Aires
  - Corporacion Medica de San Martin, San Martín, PCIA de Buenos Aires
  - Cordis - Instituto del Corazon, Resistencia, PCIA de Chaco
  - Hospital de Alta Complejidad "Pte. Juan Domingo Peron", Formosa, PCIA de Formosa
  - Hospital Provincial Dr. Jose Maria Cullen, Santa Fe, PCIA de Santa FE
  - Centro De Investigaciones Clinicas Del Litoral S.R.L., Santa Fe, PCIA de Santa FE
  - Cedir S.A - Centro De Diagnostico Y Rehabilitacion S.A., Santa Fe, PCIA de Santa FE
  - Centro Modelo de Cardiologia, San Miguel de Tucumán, PCIA de Tucuman
  - Instituto de Hematologia y Medicina Clinica "Dr. Ruben A. Davoli", Rosario, Pcia. de Santa FE
  - Instituto de Investigaciones Clinicas Rosario, Rosario, Santa Fe Province
  - Instituto Medico CENICLAR - Central de Investigaciones Clinicas Argentina -Sanatorio de la Mujer, Rosario, Santa Fe Province
  - Centro Medico CCBR Tucuman, San Miguel de Tucumán, Tucumán Province
  - Investigaciones Medicas IMOBA S.R.L., Buenos Aires
  - Universidad Maimonides, Buenos Aires
  - Centro de Investigacion: AXISMED S.R.L., Buenos Aires
  - CIPREC - Centro de Investigacion y Prevencion Cardiovascular S.A., C.a.b.a.
  - Instituto de Cardiologia y Cirugia Cardiovascular - Fundacion Favaloro, Ciudad Autonoma de B. Aires
  - Cicemo - Consultorio de Investigaciones Clinicas E.M.O. S.R.L., Ciudad Autonoma de B. Aires
  - Instituto Cardiovascular De Buenos Aires, Ciudad Autonoma de B. Aires
  - Instituto de Cardiologia de Corrientes "Juana Fca. Cabral", Corrientes
  - ILAIM Instituto Latinoamericano de Investigaciones Medicas, Córdoba
  - Clinico Chutro SRL, Córdoba
  - Centro de Investigaciones Clinicas "Instituto del Corazon", Córdoba
  - Clinica Privada Colombo, Córdoba
  - Instituto Medico DAMIC S.R.L., Córdoba
  - Centro Medico Luquez, Córdoba
  - IPAC Caraffa, Córdoba
  - Hospital Central de Mendoza, Mendoza
  - Cordis S.A., Salta
  - Centro Cardiovascular Salta, Salta
  - Instituto Cardiovascular San Luis A.E., San Luis
- Australia (29):
  - Canberra Hospital, Garran, Australian Capital Territory
  - Boden Institute of Obesity, Nutrition, Exercise and Eating Disorders, Camperdown, New South Wales
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Central Coast Neurosciences Research, Erina, New South Wales
  - Gosford Hospital, Gosford, New South Wales
  - Australian Clinical Research Network, Maroubra, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Holy Spirit Northside Private Hospital Limited, Chermside, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Core Research Group Pty Ltd, Milton, Queensland
  - Redcliffe Hospital, Redcliffe, Queensland
  - Austrials Pty Ltd, Sherwood, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - Adelaide Medical Research, Ashford, South Australia
  - SA Heart, Ashford, South Australia
  - Southern Adelaide Diabetes and Endocrine Service, Daws Park, South Australia
  - Department of Cardiology, Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Heart and Vascular Research, Fullarton, South Australia
  - Launceston General Hospital, Launceston, Tasmania
  - Eastern Health - Box Hill Hospital, Box Hill, Victoria
  - The Northern Hospital, Epping, Victoria
  - Barwon Health-The Geelong Hospital, Geelong, Victoria
  - Austin Health - Heidelberg Repatriation Hospital, Heidelberg West, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Fremantle Hospital, Fremantle, Western Australia
  - HPS Pharmacies, Joondalup, Western Australia
  - Joondalup Cardiovascular Trials Foundation Inc., Joondalup, Western Australia
  - Sir Charles Gairdner Hospital, Heart Research Institute, Nedlands, Western Australia
- Belgium (36):
  - VZW Algemeen Ziekenhuis KLINA, Brasschaat, Antwerpen
  - AZ Turnhout - campus St. Elisabeth, Turnhout, Antwerpen
  - Hopital Erasme-Universite Libre de Bruxelles (ULB), Anderlecht, Brabant Flamand
  - Centre hospitalier de Jolimont-Lobbes - Centre de Recherche Medicale de Jolimont, La Louvière, Haine Saint PAUL
  - Algemeen Stedelijk Ziekenhuis, Aalst, Oost-vlaanderen
  - Az Sint Blasius, Dendermonde, Oost-vlaanderen
  - AZ Sint Lucas Gent-Campus Sint Lucas, Ghent, Oost-vlaanderen
  - Az Glorieux, Ronse, Oost-vlaanderen
  - AZ Groeninge-Campus Loofstraat, Kortrijk, West-vlaanderen
  - Az Damiaan, Ostend, West-vlaanderen
  - A.Z. Sint-Augustinus Veurne, Veurne, West-vlaanderen
  - ZNA Campus Middelheim, Antwerp
  - Imeldaziekenhuis Bonheiden, Bonheiden
  - A.Z. St.Jan AV Brugge, Bruges
  - University Hospital Brussels - Centrum voor hart- en vaatziekten, Brussels
  - University Hospital Brussels- Diabeteskliniek, Brussels
  - Private Practice 'Cardiovascular Detection Center', De Pinte
  - ZOL Campus Sint-Jan, Genk
  - AZ Maria Middelares, Ghent
  - Grand Hopital de Charleroi, Site St-Joseph, Gilly
  - Hygeia, Hasselt
  - Jessa Ziekenhuis, Hasselt
  - Sint-Franciskusziekenhuis, Heusden-Zolder
  - Centre Hospitalier Regional de Huy, Huy
  - Jan Yperman Ziekenhuis, Cardiology, Ieper
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
  - University hospitals Leuven - Cardiology department, Leuven
  - Centre Hospitalier Chretien, Liège
  - Centre Hospitalier Universitaire de Liege, Liège
  - Huisartsenpraktijk Medilink, Linkebeek
  - Huisartsenpraktijk Luc Capiau, Massemen
  - AZ Sint-Maarten, Mechelen
  - C.H.U. Ambroise Pare, Mons
  - Mariaziekenhuis vzw, Overpelt
  - AZ Nikolaas, Sint-Niklaas
  - Dr. Luc De Wolf - Private Practice, Tienen
- Brazil (63):
  - Centro de Pesquisas em Diabetes e Doencas Endocrino-Metabolicas Ltda, Fortaleza, Ceará
  - Hospital Universitario Walter Cantidio, Fortaleza, Ceará
  - Hospital de Messejana Dr Carlos Alberto Studart Gomes, Fortaleza, Ceará
  - CEDOES - Centro de Diagnostico e Pesquisa da Osteoporose do Espirito Santo, Vitória, Espírito Santo
  - Instituto Cardiopulmonar da Bahia, Salvador, Estado de Bahia
  - Fundacao Bahiana De Cardiologia, Salvador, Estado de Bahia
  - HBA S/A ASSISTENCIA MEDICA E HOSPITALAR-Hospital da Bahia, Salvador, Estado de Bahia
  - Instituto De Cardiologia Do Distrito Federal, Brasília, Federal District
  - INGOH - Instituto Goiano de Oncologia e Hematologia, Goiânia, Goiás
  - Via Medica - Clinica Medica Integrada Ltda - Barroso e Sebba Ltda, Goiânia, Goiás
  - Liga Mineira de Ressuscitacao Cardiopulmonar, Belo Horizonte, Minas Gerais
  - Hospital Lifecenter / Lifecenter Sistema de Saude S.A, Belo Horizonte, Minas Gerais
  - Hospital Felicio Rocho, Belo Horizonte, Minas Gerais
  - Hospital Vera Cruz, Belo Horizonte, Minas Gerais
  - Hospital Universitario Ciencias Medicas / Fundacao Educacional Lucas Machado, Belo Horizonte, Minas Gerais
  - Hospital Universitário Sao José / FELUMA - MG, Belo Horizonte, Minas Gerais
  - Liga Mineira de Ressucitacao cardiopulmonar, Belo Horizonte, Minas Gerais
  - CARDSEARCH/CARDRESEARCH - Cardiologia Assistencial e de Pesquisa LTDA, Belo Horizonte, Minas Gerais
  - Universidade Federal de Uberlandia, Uberlândia, Minas Gerais
  - Eurolatino Pesquisas Medicas LTDA, Uberlândia, Minas Gerais
  - Sociedade Hospitalar Angelina Caron/Hospital e Maternidade Angelina Caron, Campina Grande do Sul, Paraná
  - Hospital Santa Casa De Curitiba, Curitiba, Paraná
  - Irmandade da Santa Casa de Misericordia de Curitiba - Hospital Santa Casa de Misericordia, Curitiba, Paraná
  - Quanta Diagnostico e Terapia / Medicina Nuclear Alto da XV, Curitiba, Paraná
  - Nucleo de Pesquisa Clínica, Curitiba, Paraná
  - Hospital Parana - Parana Medical Research Center - MARIMED SERVICOS MEDICOS S.A., Maringá, Paraná
  - Universidade Federal do Para - Hospital Universitario Joao de Barros Barreto, Belém, Pará
  - Centro de Pesquisas Medicas Basica e Clinica LTDA, Recife, Pernambuco
  - Hospital Agamenon Magalhaes, Recife, Pernambuco
  - CCBR - Centro de Pesquisas e Analises Clinicas LTDA, Rio de Janeiro, Rio de Janeiro
  - CCBR Brasil - Centro de Pesquisa e Analises Clinicas LTDA, Rio de Janeiro, Rio de Janeiro
  - Hemocardio S/S Ltda, Natal, Rio Grande do Norte
  - Hospital Universitario - Associacao Educadora Sao Carlos - AESC, Canoas, Rio Grande do Sul
  - Associacao Hospitalar Beneficente Sao Vicente de Paulo - Hospital Sao Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Santa Casa De Misericordia De Pelotas, Pelotas, Rio Grande do Sul
  - Irmandade Da Santa Casa De Misericordia De Porto Alegre - ISCMPA, Porto Alegre, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Mae de Deus/Associacao Educadora Sao Carlos AESC/IMV - Instituto de Medicina Vascular, Porto Alegre, Rio Grande do Sul
  - Uniao Brasileira de Educacao e Assistencia (UBEA) - Hospital Sao Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Hospital Santa Isabel, Blumenau, Santa Catarina
  - Insituto de Cardiologia de Santa Catarina, São José, Santa Catarina
  - Loema Medicina e Bem Estar- Centro Especializado em Cardiologia Ltda, Campinas, São Paulo
  - Scentryphar Pesquisa Clinica, Campinas, São Paulo
  - Hospital E Maternidade Celso Pierro PUC - Campinas - Sociedade Campineira de Educacao e Instrucao, Campinas, São Paulo
  - CAEP - Centro Avançado de Estudos e Pesquisas Ltda., Campinas, São Paulo
  - ICM - Instituto do Coracao de Marilia, Marília, São Paulo
  - Instituto Conceive, Paraíso, São Paulo
  - Hospital Estadual Mario Covas, Santo André, São Paulo
  - Instituto Domingo Braile _ Braile Hospital Dia LTDA, São José do Rio Preto, São Paulo
  - IMC - Instituto de Molestias Cardiovasculares/Equipamentos Cardiovasculares Rio Preto Ltda, São José do Rio Preto, São Paulo
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - CPQuali Pesquisa Clinica LTDA, São Paulo, São Paulo
  - Hospital Samaritano, São Paulo, São Paulo
  - Instituto de Conhecimento, Ensino e Pesquisa (Administrative local), São Paulo, São Paulo
  - Comed Care Empresa de Atendimento Clinico Geral - LTDA - Hospital Total Care, São Paulo, São Paulo
  - CCBR Sao Paulo, São Paulo, São Paulo
  - CEPIC - Centro Paulista de Investigacao Clinica e Servicos Medicos Ltda., São Paulo, São Paulo
  - Santa Casa de Misericordia de Votuporanga, Votuporanga, São Paulo
  - CPClin- Centro de Pesquisas Clinicas Ltda./Clinica Dr. Freddy Goldberg Eliaschewitz, São Paulo
  - FGM-Clinica Paulista de Doencas Cardiovasculares, São Paulo
  - SPDM Associacao Paulista para o Desenvolvimento da Medicina, São Paulo
  - UNIFESP - Hospital Sao Paulo - Setor de Lipides, Aterosclerose e Biologia Vascular, São Paulo
  - Instituto Jaqueline Scholz Issa e Mario Issa de Cardiologia LTDA, São Paulo
- Canada (68):
  - LMC Diabetes & Endocrinology (Calgary), Calgary, Alberta
  - Foothills Hospital/University of Calgary, Calgary, Alberta
  - Nanji Professional Corporation, Calgary, Alberta
  - The Medical Arts Health Research Group, Kelowna, British Columbia
  - Dr Stephen Pearce Inc, Surrey, British Columbia
  - Dr. Adam Yeung Inc., Surrey, British Columbia
  - Dr. Micheal Kanakos Inc, Surrey, British Columbia
  - Dr. Raymond Dong Inc., Surrey, British Columbia
  - Dr. Richard Bon Inc., Surrey, British Columbia
  - Dr. Stephen S. Cheung Inc., Surrey, British Columbia
  - SMH Cardiology Clinical Trials, Surrey, British Columbia
  - Dr Peter K.H. Tan Inc, Surrey, British Columbia
  - Dr. Dante E. Manyari Inc., Surrey, British Columbia
  - Dr. Stephanie Au, Inc., Surrey, British Columbia
  - SMH Cardiology Clinical Trials Inc., Surrey, British Columbia
  - Dr. Kapil M. Bhagirath Medical Services Corporation, Surrey, British Columbia
  - Victoria Heart Institute Foundation, Victoria, British Columbia
  - Discovery Clinical Services Ltd., Victoria, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Unicity Laboratory Services, Winnipeg, Manitoba
  - Rivergrove Medical Clinic, Winnipeg, Manitoba
  - G.A. Research Associates Ltd., Moncton, New Brunswick
  - Cardiology Research Associates of New Brunswick, Saint John, New Brunswick
  - Health Sciences Centre, St. John's, Newfoundland and Labrador
  - LMC Diabetes & Endocrinology (Brampton), Brampton, Ontario
  - Aviva Clinical Trial Group Inc., Burlington, Ontario
  - JBN Medical Diagnostic Services Inc., Burlington, Ontario
  - Philippe R. Beaudry Medicine Professional Corporation, Burlington, Ontario
  - Cambridge Cardiac Care Centre, Cambridge, Ontario
  - Vizel Cardiac Research, Saul Vizel Professional Medicine Corporation, Cambridge, Ontario
  - Moran Medical Centre, Collingwood, Ontario
  - C & L Research, Fort Erie, Ontario
  - Brian Y.L. Wong Medicine Professional Corporation, Greater Sudbury, Ontario
  - Parkdale Medical Centre, Hamilton, Ontario
  - Western University - WCPHFM, London, Ontario
  - Stroke Prevention & Atherosclerosis Research Centre (SPARC)-Siebens-Drake Research Institute, London, Ontario
  - LMC Diabetes & Endocrinology (Markham), Markham, Ontario
  - Newmarket Cardiology Research Group, Newmarket, Ontario
  - LMC Clinical Research Inc. (Oakville), Oakville, Ontario
  - LMC Oakville, Oakville, Ontario
  - The Office of Dr. James Cha, Oshawa, Ontario
  - Kawartha Cardiology Clinical Trials, Peterborough, Ontario
  - London Road Diagnostic Clinic and Medical Centre, Sarnia, Ontario
  - Sarnia Institute of Clinical Research, Sarnia, Ontario
  - Scarborough Cardiology Research Associates Inc., Scarborough Village, Ontario
  - Canadian Centre for Research on Diabetes, Smiths Falls, Ontario
  - LMC Diabetes & Endocrinology (Thornhill), Thornhill, Ontario
  - JJ Dig Research LTD, Toronto, Ontario
  - Canadian Phase Onward, Inc., Toronto, Ontario
  - LMC Diabetes & Endocrinology (Bayview), Toronto, Ontario
  - Dr. Anil K. Gupta Medicine Professional Corporation, Toronto, Ontario
  - Dr. Mohan Babapulle Medicine Professional Corporation, Waterloo, Ontario
  - Dr. Louis Yao, Weston, Ontario
  - Ecogene-21, Chicoutimi, Quebec
  - Q & T Research Chicoutimi, Chicoutimi, Quebec
  - Q&T Recherche Outaouais Inc., Gatineau, Quebec
  - Centre de Recherche Clinique de Laval, Laval, Quebec
  - Omnispec clinical research inc, Mirabel, Quebec
  - Montreal Heart Institute, Montreal, Quebec
  - Diex Research Montreal, Inc., Montreal, Quebec
  - Recherche Clinique Sigma Inc, Québec, Quebec
  - Clinique des maladies lipidiques de Quebec, Québec, Quebec
  - Centre integre de sante et de services sociaux de Lanaudiere (CISSSL), Saint-Charles-Borromée, Quebec
  - CISSS des Laurentides-Point de Service de St-Jerome- Comite d'ethique de la recherche, Saint-Jérôme, Quebec
  - St-Jerome Medical Research Inc., Saint-Jérôme, Quebec
  - LMC Diabetes & Endocrinology (Montreal), Saint-Laurent, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke- Hotel-Dieu, Sherbrooke, Quebec
  - Centre Integre de Sante et de services sociaux de Chaudiere-Appalaches (CISSS-CA), St-Georges, Beauce, Quebec
- Chile (10):
  - Corporacion de Beneficencia Osorno, Osorno, Los Lagos Region
  - Hospital Clinico Magallanes, Punta Arenas, Region de Magallanes
  - Centro de Investigacion Clínica del Sur, Temuco, Región de la Araucanía
  - Biomedica Research Group, Providencia Santiago, Santiago Metropolitan
  - CICAB, Santiago, Santiago Metropolitan
  - Servicios Medicos Godoy, Santiago, Santiago Metropolitan
  - SMOLAM, Santiago, Santiago Metropolitan
  - Hopsital y CRS El Pino, Santiago, Santiago Metropolitan
  - Complejo Asitencial Dr. Sotero del Rio, Santiago, Santiago Metropolitan
  - Quantum Research, Puerto Varas
- China (30):
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Haikou People's Hospital, Haikou, Hainan
  - The 2nd Affiliated Hospital Of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Habrin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital Of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital Of Zhengzhou University, Zhengzhou, Henan
  - The Central Hospital Of Wuhan, Wuhan, Hubei
  - Pu Ai Hospital of Wuhan City, Wuhan, Hubei
  - Changde First People's Hospital, Changde, Hunan
  - Changsha Central Hospital, Changsha, Hunan
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - Xiangtan City Central Hospital, Xiangtan, Hunan
  - Zhuzhou Central Hospital, Zhuzhou, Hunan
  - Inner Mongolia Baogang Hospital, Baotou, Inner Mongolia
  - Inner Mongolia Autonomous Region People's Hospital, Hohhot, Inner Mongolia
  - Wuxi People's Hospital, Jiangsu, Jiangsu
  - Suzhou Kowloon Hospital Shanghai Jiaotong University School of Medicine, Suzhou, Jiangsu
  - The affiliated Hospital of Xuzhou Medical College, Xuzhou, Jiangsu
  - Jilin Province People's Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - General Hospital Of Ningxia Medical University, Yinchuan, Ningxia
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - The First Affiliated Hospital Of Xinjiang Medical University, Ürümqi, Xinjiang
  - Ningbo First hospital, Ningbo, Zhejiang
  - Beijing Chao-yang Hospital, Beijing
  - FuWai Hospital, CAMS & PUMC, Beijing
  - Shanghai General Hospital, Shanghai
  - Tianjin Union Medical Center, Tianjin
  - Taizhou Hospital of Zhejiang Province, Zhejiang
- Colombia (22):
  - Hospital Pablo Tobon Uribe, Medellín, Antioquia
  - Centro de Investigacion Clinica Avanzada y Multidisciplinaria CICLAM, Medellín, Antioquia
  - Centro de Medicina del Ejercicio y Rehabilitacion Cardiac - CEMDE S.A., Medellín, Antioquia
  - Rodrigo Botero S.A.S., Medellín, Antioquia
  - Clinica De La Costa Ltda, Barranquilla, Atlántico
  - Centro Cientifico Asistencial Jose Luis Accini S.A.S., Barranquilla, Atlántico
  - Corazon Ips Sas., Barranquilla, Atlántico
  - Fundacion del Caribe Para La Investigacion Biomedica - Fundacion BIOS, Barranquilla, Atlántico
  - Asociacion IPS Medicos Internistas de Caldas, Manizales, Caldas Department
  - Hospital Universitario San Ignacio, Bogota D C, Cundinamarca
  - MedPlus Medicina Prepagada S.A., Bogota D.C., Cundinamarca
  - Instituto de Investigacion Endocrinologia y Prevencion Metabolica - ENDOCARE LTDA., Bogota D.C., Cundinamarca
  - Simedics Ips Sas, Bogota D.C., Cundinamarca
  - Solano & Terront Servicios Medicos Ltda-Establecimiento Comercial UNIENDO, Bogota D.C., Cundinamarca
  - Dexadiab Servicios Medicos LTDA, Bogota D.C, Cundinamarca
  - Caja de Compensacion Familiar CAFAM, Sede Centro de Atencion en Salud CAFAM FLORESTA, Bogota D.C, Cundinamarca
  - Healthy Medical Center S.A.S, Zipaquirá, Cundinamarca
  - Centro de Diagnostico Cardiologico LTDA., Cartagena, Departamento de Bolívar
  - Fundacion Centro de Obesidad y Metabolismo COMETA, Pasto, Departamento de Nariño
  - Instituto del Corazon de Bucaramanga S.A., Bucaramanga, Santander Department
  - Fundacion Cardiovascular De Colombia - Instituto del Corazón Floridablanca, Floridablanca, Santander Department
  - Fundacion Reina Isabel, Cali, Valle del Cauca Department
- Czechia (28):
  - Edumed S.R.O., Broumov, Královéhradecký kraj
  - EDUMED s.r.o., Jaroměř, Královéhradecký kraj
  - Kardiologicka ambulance, Trutnov, Královéhradecký kraj
  - Lekarna na Poliklinice, Trutnov, Královéhradecký kraj
  - Mudr. Jan Vrkoc S.R.O., Ostrava, Moravskoslezský kraj
  - Pv-Kardiologie S.R.O., Pardubice, Pardubický kraj
  - Kardiologicka Ambulance, Brno, South Moravian
  - CCBR Czech Brno, s.r.o., Brno
  - DIKa centrum s.r.o., Kardiologicka a interni ambulance, Havířov
  - Fakultni Nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fremlova Apotheca s.r.o., Litovel
  - Kardio interna s.r.o., Litovel
  - Fakultni Nemocnice Olomouc, Olomouc
  - CCBR Czech a.s., Pardubice
  - Kardiologie Plzen s.r.o., Pilsen
  - Fakultni Nemocnice Kralovske Vinohrady, Prague
  - Fakultni poliklinika Vseobecne fakultni nemocnice v Praze, Prague
  - CCBR Czech Prague, s.r.o, Prague
  - Centrum kardiovaskularni prevence 1. LF UK a TN, Prague
  - Kardiologie a interni lekarstvi, Prague
  - NEFROMED, s.r.o., Prague
  - Interna a kardiologie s.r.o., Rožnov pod Radhoštěm
  - Nemocnice Pardubickeho kraje, a.s., Svitavska nemocnice, Svitavy
  - Ordinace V Tabacce s.r.o., Tábor
  - MUDr. Antonin Dufka, kardiologicka ambulance, Uherské Hradiště
  - MUDr. Nina Zemkova s.r.o., Uherské Hradiště
  - KIGE s.r.o., Znojmo
- Denmark (26):
  - Aabenraa Hospital Hjertemedicinsk klinik Kredslobscentret, SHS, Aabenraa
  - Sygehus Sonderjylland Aabenraa, Aabenraa
  - Aalborg Universitetshospital, Lipidklinikken, Aalborg
  - CCBR Aalborg, Aalborg
  - Aarhus Universitetshospital Skejby, Hjertesygdomme ¿ Klinisk Forskning, Aarhus
  - CCBR Ballerup, Ballerup Municipality
  - Bispebjerg og Frederiksberg Hospital, Copenhagen NV
  - Sydvestjysk Sygehus, Hjertemedicinsk Projektgruppe, Esbjerg
  - Frederiksberg Hospital, Frederiksberg
  - Glostrup Hospital, Glostrup Municipality
  - Herlev Universitetshospital, Herlev
  - Regionshospitalet Herning, Herning
  - Hillerod Hospital, Hillerød
  - Hvidovre Universitetshospital, Hvidovre
  - Region Sjaelland Sygehus Nord, Koge Sygehus, Koege
  - Kolding Sygehus, Kolding
  - Amager Hospital, København S
  - Karkirurgisk Klinisk, København Ø
  - Nykobing F. Sygehus-Medicinsk afdeling, Nykøbing Falster
  - Region Sjaelland Naestved Sygehus, Næstved
  - Regionshospitalet Randers, Randers
  - Regionshospitalet Silkeborg, Hjerte Projektkontor, Silkeborg
  - Slagelse Sygehus, Slagelse
  - Svendborg Sygehus, Svendborg
  - CCBR Vejle, Vejle
  - Hospitalsenheden Midt, Regionshospital Viborg, Viborg
- Finland (23):
  - HYKS Jorvin sairaala, Espoo
  - Linnan Klinikka Oy, Hämeenlinna
  - Geri-Med Oy, Helsinki
  - Helsinki University Central Hospital, Helsinki
  - Helsingin yliopistollinen keskussairaala, Sisaetaudit ja kuntoutus, Biomedicum 2U, Helsinki
  - Ita-Suomen laakarikeskus Oy, Joensuu
  - StudyCor Oy, Jyväskylä
  - Laeaekaerikeskus Aava Kerava, Kerava
  - Menoa oy, Kinkomaa
  - Kokkolan Keskussairaala, Kokkola
  - Mewell liikuntaklinikka, Kotka
  - Itae-Suomen Laeaekaeritalo, Kuopio
  - Terveystalo Kuopio, Kuopio
  - Oulu Mentalcare Oy, Oulu
  - Terveystalo Oulu, Diapolis, Oulu
  - Oulu University Hospital, Oulu
  - Porin Laakaritalo Oy, Pori
  - Terveystalo Siilinjarvi, Siilinjärvi
  - FinnMedi Oy, Tampere
  - Terveystalo Pulssi, Turku
  - Turku University hospital, Turku
  - Vantaan Tutkimuskeskus, Vantaa
  - Ylitornion Terveyskeskus, Ylitornio
- France (21):
  - CHU Jean Minjoz Cardiologie, Besançon
  - Groupe Hospitalier de Pellegrin Hopital Pellegrin, Bordeaux
  - Centre Hospitalier De Bourg En Bresse - Hopital Fleyriat, Bourg-en-Bresse
  - centre hospitalier Sub-Francilien, Corbeil-Essonnes
  - Scp Cardiovasculaire De L'Est, Essey-lès-Nancy
  - Centre Hospitalier Louis Pasteur, Le Coudray
  - Hopital La Louviere, Lille
  - Centre Hospitalier Saint Philibert, Lomme
  - Hopital Cardiovasculaire Et Pneumologique Louis Pradel, Lyon
  - Hopital Arnaud de Villeneuve - CHU Montpellier, Montpellier
  - CHU de Nantes - Hopital Nord Laennec, Nantes
  - Nouvelles Cliniques Nantaises, Nantes
  - Chu De Nice - Hopital Pasteur, Nice
  - Hopital Cardiologique, Pessac
  - CHU de Poitiers, Poitiers
  - CHU de Renes Hopital de Pontchaillou, Rennes
  - CHU de Toulouse, Toulouse
  - Hospital Cuy Chatilliez, Tourcoing
  - Hopital Trousseau, Tours
  - Centre Hospitalier (GH) de Valenciennes, Valenciennes
  - Polyclinique Vauban, Valenciennes
- Germany (70):
  - Universitaets Herzzentrum Freiburg Bad Krozingen, Bad Krozingen, Baden-Wurttemberg
  - Medizinische Universitaetsklinik Heidelberg, Heidelberg, Baden-Wurttemberg
  - Gemeinschaftspraxis im Altstadt Carree, Fulda, Hesse
  - Zentrum Klinische Studien Neuwied (ZKSN), Neuwied, Rhineland-Palatinate
  - Gemeinschaftspraxis Schwabenheim, Schwabenheim, Rhineland-Palatinate
  - Klinikum Altenburger Land Gmbh, Altenburg
  - Forschungszentrum Dr. med Irma Schoell, Bad Homburg
  - Institut fuer Klinische Forschung und Entwicklung(IKFE) Berlin GmbH, Berlin
  - Klinische Forschung Berlin- Mittte GmbH, Berlin
  - POLIKUM Institut GmbH, Polikum Berlin Friedenau, Berlin
  - DRK Kliniken Berlin Kopenick, Zentrum Klinische Forschung, Berlin
  - Synexus Clinical Research GmbH, Berlin
  - Deutsches Herzzentrum Berlin, Berlin
  - Medizinisches Versorgungszentrum am Bahnhof Spandau, Berlin
  - Staedtische Kliniken Bielefeld Gem. GmbH - Klinikum Mitte, Bielefeld
  - Bochum Research Centre-Synexus Clinical Research GmbH, Bochum
  - Synexus Clinical Research GmbH, Bochum
  - MediClin Reha-Zentrum Spreewald, Burg
  - Klinikum Coburg, Coburg
  - Zentrum fuer klinische Forschung, Cologne
  - Kardiologische Praxisgemeinschaft, Dortmund
  - St. Johannes-Hospital, Dortmund
  - Gemeinschaftspraxis fuer Kardiologie Dres. Med. Willgeroth/Wetzel, Dortmund
  - Klinsche Forschung Dresden GmbH, Dresden
  - Praxis Dr. med. Christoph Axthelm, Dresden
  - GWT-TUD GmbH, Studienzentrum Professor Hanefeld, Dresden
  - Gemeinschaftspraxis Dr. Hagemann/Breiderhoff/Durfeld, Essen
  - Medizentrum Essen Borbeck, Essen
  - Studienzentrum, Essen
  - Gemeinschaftspraxis Dres. Dirk Weber, Ulrich Weber, Heiner Saueressig, Birte Turner und Georg, Essen
  - Schwerpunktpraxis Dr. Luedemann fuer Diabetes Gefaess- und Ernaehrungsmedizin, Falkensee
  - Synexus Clinical Research GmbH, Frankfurt
  - Clinphenomics Gmbh & Co Kg, Studienzentrum, Frankfurt
  - IKF Institut fuer klinische Forschung Frankfurt, Frankfurt am Main
  - Klinik und Poliklinik fuer Innere Medizin B - Kardiologie, Angiologie, Pulmologie, Greifswald
  - Cardiologicum Hamburg, Hamburg
  - Praxis Dr. med Cornelia Brauer, Hamburg
  - Klinische Forschung Hannover-Mitte GmbH, Hanover
  - Universitaetsklinikum des Saarlandes Klinik fuer Innere Medizin III, Homburg
  - Praxis Dr. Heister, Kamp-Lintfort
  - Studienzentrum Dr. Appel, Kassel
  - Gemeinschaftspraxis Dr. Klein / Minnich, Künzing
  - Klinik fur Innere Medizin, Kardiologie und Angiologie MediClin Herzzentrum Lahr/Baden., Lahr
  - Synexus Leipzig Clinical Research Centre, Leipzig
  - SIBAmed Studienzentrum GmbH & Co. KGKG, Leipzig
  - Gemeinschaftspraxis Dr. med. Heidrun Taeschner und Dr. med. Susanne Bonigut, Leipzig
  - Klinikum Leverkusen GgmbH, Leverkusen
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH, Ludwigshafen
  - Maerkische Kliniken GmbH, Klinikum Luedenscheid, Innere III, Lüdenscheid
  - Klinikum Lunen, St. Marienhospital, Lünen
  - SMO.MD GmbH, Zentrum fuer klinische Studien Site Management and Clinical Research Unit, Magdeburg
  - Pfuetzner Science & Health Institute-Gmbh, Mainz
  - Ze:ro Arztpraxen Dr. med. Salbach, Mannheim
  - Klinikum Fur Herz- & Kreislauferkrankungen, Munich
  - Staedtisches Klinikum Muenchen GmbH, Klinikum Neuperlach, Munich
  - Klinikum Der Universitat Munchen, München
  - Klinikum fuer Herz- & Kreislauferkrankungen, München
  - Kardiologische Praxis Northeim, Northeim
  - Gemeinschaftspraxis Drs Haggenmiller/Jeserich, Kardiologie, Angiologie, Innere Medizin, Nuremberg
  - Allgemeinmedizinisch-Internistische Praxisgemeinschaft, Offenbach
  - Praxis Dres. Med Naudts und Nowack, Rodgau
  - Klinik Am See - Klinik Am See - Rehabilitationszentrum Fur Innere Medizin, Rüdersdorf
  - Klinische Forschung Schwerin GmbH, Schwerin
  - Kardiologische Gemeinschaftspraxis Dres Med. Gerke/Buerger, Soest
  - Praxisgemeinschaft Stuhr-Brinkum, Stuhr-Brinkum
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Universitaetsklinikum Ulm, Ulm
  - Josephs-Hospital Warendorf Med. Klinik II, Kardiologie/Angiologie, Warendorf
  - Kardiologische Praxis, Wermsdorf
  - ForschungszentrumRuhr KliFoCenter GmbH, Witten
- Hungary (32):
  - Pecsi Tudomanyegyetem AOK, II., Pécs, Baranya
  - Bacs-Kiskun Megyei Korhaz, Kecskemét, Bács-Kiskun county
  - Szegedi Tudomanyegyetem AOK, I. sz Belgyogyaszati Klinika, Szeged, Csongrád megye
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár, Fejér
  - DRC Kft., Balatonfüred
  - DRC Kft., Balatongyörök
  - Grof Tisza Istvan Korhaz Berettyoujfalu, Berettyóújfalu
  - Kardiologiai Maganrendelo, Békéscsaba
  - Budapesti Szent Ferenc Korhaz, Budapest
  - Synexus Magyarorszag Kft, Budapest
  - Szent Rokus Korhaz, Budapest
  - Semmelweis Egyetem, Budapest
  - Gottsegen Gyorgy Orszagos Kardiologiai Intezet, Budapest
  - Egyesitett Szent Istvan es Szent Laszlo Korhaz-Rendelointezet, Budapest
  - Bajcsy-Zsilinszky Korhaz es Rendelointezet, Budapest
  - Szent Janos Korhaz es Eszak-budai Egyesitett Korhazak, III. Belgyogyaszat-Kardiologiai Osztaly, Budapest
  - Debreceni Egyetem, I. sz. Belgyogyaszati Klinika, Debrecen
  - Synexus Magyarorszag Egeszsegugyi Szolgaltato Kft., Debrecen
  - Synexus Magyarorszag Kft., Gyula
  - Edes Szivunk Egeszsegkozpont Kft., Hajdúszoboszló
  - BKS Research Kft., Albert Schweitzer Korhaz, Hatvan
  - Somogy Megyei Kaposi Mór Oktató Kórház, Kaposvár
  - Jutrix Egeszsegugyi Kft, Kecskemét
  - Pest Megyei Flor ferenc Korhaz, Kistarcsa
  - Josa Andras Oktatokorhaz, Nyíregyháza
  - Medifarma-98 Kft., Nyíregyháza
  - Pecsi Tudomanyegyetem AOK, I. Belgyogyaszati Klinika, Pécs
  - Mentahaz Maganorvosi Kozpont, Székesfehérvár
  - Hetenyi Geza Korhaz, Szolnok
  - Markusovszky Egyetemi Oktatokarhaz, Szombathely
  - Dr. Sydo es Tsa Kft, Veszprém
  - Zala Megyei Korhaz, Zalaegerszeg
- India (12):
  - Dr. Jivraj Mehta Smarak Health Foundation, Bakeri Medical Research Centre, Ahmedabad, Gujarat
  - Apex Heart Institute (A Unit of TCVS Pvt. Ltd), Ahmedabad, Gujarat
  - SAL Hospital, Ahmedabad, Gujarat
  - Apple Hospital, Surat, Gujarat
  - Unicare Heart Institute & Research Center, Surat, Gujarat
  - BAPS - Pramukh Swami Hospital, Surat, Gujarat
  - Rhythm Heart Institute, Vadodara, Gujarat
  - Aster Aadhar Hospital (Prerana Hospital Ltd.), Kolhāpur, Maharashtra
  - Shri Krishna Hrudayalaya and Critical Care Centre, Nagpur, Maharashtra
  - Jehangir Clinical Development Centre Pvt. Ltd., Pune, Maharashtra
  - Mediciti Hospitals, Hyderabad, Telangana
  - M.V. Hospital And Research Centre, Lucknow, Uttar Pradesh
- Ireland (6):
  - Beaumont Hospital, Dublin, Leinster
  - The Adelaide & Meath Hospital-Dublin Incorporating The National Children's Hospital, Dublin
  - Mater Misericordiae University Hospital, Dublin
  - St. James's Hospital, Dublin
  - Health Research Board, Galway
  - Portiuncula Hospital, Galway
- Israel (25):
  - Barzilai Medical Center, Ashkelon
  - Gefen Institute for Research and Cardiac Health, Bat Yam
  - The Soroka University Medical Center, Beersheba
  - Ben Yair Community Clinic - Clalit Health Services, Beersheba
  - Heart Institute, Hillel Yaffe Medical Center, Hadera
  - Rambam Medical Center, Haifa
  - Cardiovascular Clinical Research Institute, Haifa
  - Edith Wolfson Medical Center, Holon
  - Heart Institute, Bikur Cholim Campus, Shaare Zedek Medical Center, Jerusalem
  - Hadassah Ein Kerem Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Galilee Medical Center, Cardiology Department, Nahariya
  - E.M.M.S Nazareth Hospital, Nazareth
  - Rabin Medical Center, Beilinson Hospital, Petah Tikva
  - Rabin Medical Center-Beilinson Hospital, Petah Tikva
  - Rabin Medical Center, Petah Tikva
  - Sha'aria Clinic, Clalit Health Services, Petah Tikva
  - Shuali Community Clinic, Clalit Health Services, Raanana
  - Department of Neurology & Sagol Neuroscience Center, Ramat Gan
  - Heart Institute, Kaplan Medical Center, Rehovot
  - Kaplan Medical Center, Rehovot
  - Internal Medicine A, Ziv Medical Center, Safed
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Assuta Medical Center, Tel Aviv
  - The Chaim Sheba Medical Center, Tel Litwinsky
- Italy (26):
  - A.O. Treviglio e Caravaggio, Treviglio (BG), Bergamo
  - AOU Policlinico "Mater Domini" UOC di Medicina interna, Catanzaro, CZ
  - Ospedale S. L. Mandic di Merate, Merate, Lecco
  - IRCCS Centro Cardiologico Fondazione Monzino, Milan, MI
  - Ospedale Civile Di Piove Di Sacco, Piove di Sacco, Padova
  - AOU Policlinico "P. Giaccone" Dipartimento delle Patologie Emergenti, Unita di Medicina Interna, Palermo, PA
  - Ospedale S. Maria della Misericordia Dipartimento di Medicina, Medicina Interna,, Perugia, PG
  - Azienda Ospedaliera Della Provincia Di Lecco - Ospedale Manzoni, Lecco, Province OF Lecco
  - Dept."Medicina lnterna e Specialita Mediche" dell' Universita degli, Roma, RM
  - Policlinico Umberto I di Roma, Rome, RM
  - Azienda Ospedaliera S'Andrea di Roma - UOC Cardiologia, Rome, RM
  - Presidioospedaliero di san dona 'di PIAVE, San Dona Di Paive, Venezia
  - Ospedale G. Fracastoro, San Bonifacio, Verona
  - AOUI di Verona - Ospedale Civile Maggiore Borgo Trento, Verona, VR
  - I.N.R.C.A. di Ancona Ospedale Geriatrico, Ancona
  - Ospedale Civile Regionale San Martino, Belluno, Belluno
  - Azienda Ospedaliera G. Brotzu, Cagliari
  - Divisione di Cardiologia con UTIC ed Emodinamica, Naples
  - Department of Clinical Medicines and Cardiovascular Sciences, Universita "Federico II" di Napoli, Napoli
  - Divisione di Cardiologia con Utic ed Emodinamica - AOU Federico II di Napoli, Napoli
  - A.O. di Reggio Emilia Arcispedale "S. Maria Nuova"/IRCCS, Reggio Emilia
  - AUSL Della Romagna-Ospedale Infermi, Rimini
  - Policlinico Umberto I di Roma - DAI Malattie Cardiovascolari e Respiratorie, Rome
  - Ospedale Santa Maria della Misericordia Azienda ULSS 18 of Rovigo, Rovigo
  - A.O.U. San Giovanni di Dio e Ruggi d'Aragona U.O.C. UTIC, Salerno
  - Azienda Ospedaliera Universitaria Santa Maria Della Misericordia, Udine
- Mexico (47):
  - Consultorio Dr. Leocadio Gerardo Munoz Beltran, Cd. Juarez, Chihuahua
  - Centro Especializado En Diabetes, Obesidad Y Prevencion De Enfermedades Cardiovasculares, S.C., México, D F
  - Centro de Investigacion Clinica del Pacifico, S.A. de C.V., Acapulco de Juárez, Guerrero
  - Investigacion Biomedica Aplicada de Hidalgo S.A. de C.V., Pachuca, Hidalgo
  - Centro de Investigacion Medica Integral S.C., Guadalajara, Jalisco
  - Instituto de Terapeutica Experimental y Clinica (INTEC) Centro Universitario de Ciencias de la Salud, Guadalajara, Jalisco
  - Hospital Mexico Americano S.C. (Emergencies), Guadalajara, Jalisco
  - Consultorio Privado del Dr. Gabriel Arturo Ramos Lopez, Guadalajara, Jalisco
  - CICEJ Centro de Investigacion Clinica Endocrinologica de Jalisco SC, Guadalajara, Jalisco
  - Unidad de Investigacion Clinica y Atencion Medica HEPA S.C., Guadalajara, Jalisco
  - Jardines Hospital de Especialidades S.A de C.V, Zapopan, Jalisco
  - Centro de Atencion e Investigacion en Factores de Riesgo Cardiovascular Omega S.C, Mexico City, Mexico City
  - Consultorio de Endocrinologia y Nutriologia, Mexico City, Mexico City
  - Operadora de Hospitales Angeles S.A. de C.V.(Emergencies), Mexico City, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion "Salvador Zubiran", Mexico City, Mexico City
  - Instituto de Diabetes Obesidad y Nutricion, S.C., Cuernavaca, Morelos
  - Hospital Inovamed Cuernavaca (Emergencies), Cuernavaca, Morelos
  - Accelerium S. de R.L. de C.V., Monterrey, Nuevo León
  - Hospital y Clinica OCA, S.A. de C.V., Monterrey, Nuevo León
  - Monterrey International Research Center, Monterrey, Nuevo León
  - Cardiolink Clin Trials, S.C., Monterrey, Nuevo León
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - Hospital Universitario De Monterrey- "Doctor Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - CRI Centro Regiomontano de Investigacion SC, Monterrey, Nuevo León
  - Global Trial Research Center S.A. de C.V., Monterrey, Nuevo León
  - Fundacion Santos y de la Garza Evia I.B.P. (Centro Medico Zambrano Hellion), San Pedro Garza García, Nuevo León
  - Centro Integral Medico SJR S.C, San Juan del Río, Querétaro
  - Centro para el Desarrollo de la Medicina y de Asistencia Médica Especializada S.C., Culiacán, Sinaloa
  - Hospital Angeles Culiacan (Emergencies Only), Culiacán, Sinaloa
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares S.C., Tampico, Tamaulipas
  - Centro de Especialidades Medicas del Estado de Veracruz, Xalapa, Veracruz
  - Instituto Biomedico De Investigacion A.C., Aguascalientes
  - Centro de Investigacion Cardiometabolica de Aguascalientes S.A. de C.V., Aguascalientes
  - Centro Hospitalario Mac, S.A. de C.V. (Emergencies), Aguascalientes
  - Hospital Cardiologica Aguescalientes, Aguascalientes
  - Unidad de Investigacion en Salud de Chihuahua S.C., Chihuahua City
  - Investigacion en Salud y Metabolismo S.C., Chihuahua City
  - Consultorio Medico de Especialidad Dr. Demetrio Kosturakis Garcia, Chihuahua City
  - Investigacion en Salud y Metabolismo S.C, Chihuahua City
  - Instituto Nacional de Ciencia Medicas y Nutricion Salvador Zubiran, Distrito Federal
  - Lahoja Asociacion para la Investigacion y Farmacovigilancia S.C., Durango
  - Cardioprevent, S.C., Durango
  - Pharmacology and Clinical Research S.A. de C.V., Querétaro
  - Cardioarritmias e Investigacion S.C., San Luis Potosí City
  - Hospital Lomas de San Luis Intemacional (Emergencies), San Luis Potosí City
  - "Hospital Central ""Dr. Ignacio Morones Prieto""", San Luis Potosí City
  - Centro Especializado En Diabetes Y Metabolismo, Veracruz
- Netherlands (71):
  - Zuyderland MC, Sittard-Geleen, Limburg
  - Isala, Zwolle, Overijssel
  - Tjongerschans Ziekenhuis, Heerenveen, Provincie Friesland
  - St. Franciscus Gasthuis, Rotterdam, South Holland
  - Het Lange Land Ziekenhuis, Zoetermeer, South Holland
  - Noordwest Ziekenhuisgroep, Alkmaar
  - EB Flevoresearch, Almere Stad
  - Meander Medical Center, Amersfoort
  - Meander Medisch Centrum, Amersfoort
  - Amstelland Hospital, Amstelveen
  - Bovenij Ziekenhuis, Amsterdam
  - OLVG, locatie West, Amsterdam
  - VU University Medical Center, Amsterdam
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Academic Medical Center, Amsterdam
  - Gelre Hospitals, Apeldoorn
  - Rode Kruis Ziekenhuis, Beverwijk
  - Tergooi Ziekenhuis, Blaricum
  - Andro Medical Research B.V., Breda
  - Amphia Ziekenhuis, Breda
  - Reinier de Graaf ziekenhuis, Delft
  - Deventer Ziekenhuis, Deventer
  - Van Weel Bethesda Hospital, Dirksland
  - Slingeland Ziekenhuis, Doetinchem
  - Albert Schweitzer Hospital, Dordrecht
  - Ziekenhuis Gelderse Vallei, Ede
  - Andromed Eindhoven, Eindhoven
  - Heartcentre Catharina Hospital, Eindhoven
  - Medisch Spectrum Twente, Enschede
  - Beatrix Ziekenhuis, Gorinchem
  - Groene Hart Ziekenhuis, Gouda
  - University Medical Center Groningen, Groningen
  - Martini Ziekenhuis, Groningen
  - Spaarne Gasthuis, Haarlem
  - St. Jansdal Ziekenhuis, Harderwijk
  - Zuyderland Medisch Centrum, Heerlen
  - Zuyderland, Heerlen
  - Treant Zorggroep, location Bethesda, Hoogeveen
  - Vascular Research Centre, Hoorn
  - Quality Care Research, Kloosterhaar
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Leiden University Medical Center, Leiden
  - Alrijne Ziekenhuis, Leiden
  - Alrijne Ziekenhuis, Leiderdorp
  - GCM Maarssenbroek, Maarssen
  - Maastricht University Medical Center, Maastricht
  - Isala Diaconessenhuis, Meppel
  - St Antonius Hospital, Nieuwegein
  - Radboud University Nijmegen Medical Centre, Nijmegen
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Waterland Hospital, Purmerend
  - Andro Medical Research B.V, Rotterdam
  - Rotterdam Research Institute, Rotterdam
  - St. Fransiscus Gasthuis, Rotterdam
  - Ikazia Ziekenhuis, Rotterdam
  - D&A Research and Genetics, Sneek
  - Hedramed, The Hague
  - Hagaziekenhuis, The Hague
  - HMC (Haaglanden Medisch Centrum) Bronovo, The Hague
  - Ziekenhuis Rivierenland, Tiel
  - Elisabeth-TweeSteden Ziekenhuis (previously named St. Elisabeth Ziekenhuis), Tilburg
  - St. Elisabeth Ziekenhuis, Tilburg
  - Elisabeth TweeSteden Ziekenhuis (ETZ), Tilburg
  - Bernhoven Ziekenhuis, Uden
  - EB Utrecht, Utrecht
  - Universitair Medisch Centrum (UMC) Utrecht - Locatie AZU, Utrecht
  - University Medical Center Utrecht, Utrecht
  - Maxima Medisch Centrum, Veldhoven
  - VieCuri Medisch Centrum, Venlo
  - Twee Steden Ziekenhuis, Waalwijk
  - Albert Schweitzer Hospital, Zwijndrecht
- New Zealand (17):
  - Optimal Clinical Trials, Grafton, Auckland
  - Henderson Medical Centre, Henderson, Auckland
  - Middlemore Hospital, Otahuhu, Auckland
  - North Shore Hospital, Takapuna, Auckland
  - Hawke's Bay Hospital, Frimley, Hastings
  - Auckland City Hospital, Auckland
  - Lipid and Diabetes Research Group, Christchurch
  - Southern Clinical Trials Shirley Ltd, Christchurch
  - Southern Clinical Trials Riccarton, Christchurch
  - RMC Medical Research Ltd., Dunedin
  - Taranaki Base Hospital, New Plymouth
  - Rotorua Hospital, Rotorua
  - Clinical Horizons NZ Ltd., Tauranga
  - Clinical Trials Unit,Bay of Plenty(BOP) Clinicla School, Tauranga
  - Papamoa Pines Medical Centre, Tauranga
  - Clinical Horizons NZ Ltd, Tauranga
  - Wellington Hospital, Wellington
- Poland (81):
  - Synexus Polska Sp. z o.o Oddzial w Poznaniu, Poznan, Greater Poland Voivodeship
  - Nzoz "Twoja Przychodnia", Poznan, Greater Poland Voivodeship
  - NZOZ Vitamed, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Nzoz Centrum Medyczne Kermed, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Specjalistyczna Praktyka Lekarska Piotr Kubalski, Grudziądz, Kuyavian-Pomeranian Voivodeship
  - Specjalistyczne Gabinety Lekarskie "Medicor Plus" - Jerzy Kopaczewski, Włocławek, Kuyavian-Pomeranian Voivodeship
  - Landa Specjalistyczne Gabinety Lekarskie, Krakow, Lesser Poland Voivodeship
  - Krakowski Szpital Specjalistyczny im. Jana Pawla II, Krakow, Lesser Poland Voivodeship
  - Szpital Specjalistyczny im. J. Dietla w Krakowie, Oddzial Kardiologii, Krakow, Lesser Poland Voivodeship
  - Centrum Medyczne Zdrowa J. Trebacz, W. Zajdel Spolka jawna, Krakow, Lesser Poland Voivodeship
  - CENTRUM MEDYCZNE A-Z Clinic, Krakow, Lesser Poland Voivodeship
  - Krakowskie Centrum Medyczne Sp. z o.o., Krakow, Lesser Poland Voivodeship
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Szpital Uniwersytecki w Krakowie,, Krakow, Lesser Poland Voivodeship
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Szpital Uniwersytecki W Krakowie, Ambulatoria, Krakow, Lesser Poland Voivodeship
  - NZOZ Centrum Zdrowia i Profilaktyki Dabie Sp. z.o.o., Krakow, Lesser Poland Voivodeship
  - Niepubliczny Zaklad Opieki Zdrowotnej Centrum Medyczne ProMiMed sp z o.o., sp.k., Krakow, Lesser Poland Voivodeship
  - NeuroCor Banaszkiewicz, Kulaga, Ostrowska, Tomaszewski lekarze spolka partnerska, Myślenice, Lesser Poland Voivodeship
  - INTERCARD Sp. z. o. o. Centrum Kardiologii Inwazyjnej, Elektroterapii i Angiologii w Nowym Targu, Nowy Targ, Lesser Poland Voivodeship
  - Medicome Sp. z o.o., Oświęcim, Lesser Poland Voivodeship
  - Centrum Szybkiej Diagnostyki Kardiologicznej Kardiomed M. Zabowka E. Zabowka, Tarnów, Lesser Poland Voivodeship
  - Specjalistyczny Gabinet Lekarski Internistyczno-Kardiologiczny Boguslaw Derlaga, Tarnów, Lesser Poland Voivodeship
  - Jeleniogorskie Centrum Chorob Serca, Przychodnia Kardiologiczna, Poradnia Kardiologiczna, Jelenia Góra, Lower Silesian Voivodeship
  - Zdrowie s.c. Agnieszka i Donald Drozdz, Wroclaw, Lower Silesian Voivodeship
  - Halina Serafin NZOZ Centrum Medyczne SERAFIN-MED, Żarów, Lower Silesian Voivodeship
  - Clinical Best Solutions, Lublin, Lublin Voivodeship
  - Optimamed Specjalistyczne Gabinety Lekarskie, Lublin, Lublin Voivodeship
  - KO-MED Centra Kliniczne Lublin II, Lublin, Lublin Voivodeship
  - KO-MED Centra Kliniczne Pulawy, Puławy, Lublin Voivodeship
  - KO-MED Centra Kliniczne Zamosc, Zamość, Lublin Voivodeship
  - Synexus Polska Sp. z o.o. Oddzial w Katowicach, Katowice, Masovian Voivodeship
  - Niepubliczny Zaklad Opieki Zdrowotnej Specjalistyczna Przychodnia Lekarska "MEDIKARD", Płock, Masovian Voivodeship
  - Centrum Medyczne Piaski Filia nr 9, Warsaw, Masovian Voivodeship
  - Instytut Kardiologii im. Prymasa Tysiaclecia Stefana Kardynala Wyszynskiego, Warsaw, Masovian Voivodeship
  - Wojskowy Instytut Medyczny,Centralny Szpital Kliniczny Ministerstwa Obronty Narodowej, Warsaw, Masovian Voivodeship
  - Instytut Kardiologii im, Warsaw, Masovian Voivodeship
  - Specjalistyczny Osrodek Medycyny Wieku Dojrzalego Sp. z o.o., Warsaw, Masovian Voivodeship
  - Szpital Specjalistyczny w Brzozowie, Podkarpacki Osrodek Onkologiczny im. Ks. B. Markiewicza Oddzial, Brzozów, Podkarpackie Voivodeship
  - INTERCARD Sp. z o.o. Centrum Kardiologii Inwazyjnej, Elektroterapii i Angiologii w Krosnie, Krosno, Podkarpackie Voivodeship
  - EMED Centrum Uslug Medycznych Ewa Smialek, Rzeszów, Podkarpackie Voivodeship
  - "OSTEO-MEDIC" s.c. Artur Racewicz, Jerzy Supronik, Bialystok, Podlaskie Voivodeship
  - Podlaski Osrodek Kardiologii Janusz Korecki, Bialystok, Podlaskie Voivodeship
  - Synexus Polska Sp. z o.o. Oddzial w Gdansku, Gdansk, Pomeranian Voivodeship
  - Niepubliczny Zaklad Opieki Zdrowotnej Gdanskie Centrum Zdrowia, Poradnia Kardiologiczna, Gdansk, Pomeranian Voivodeship
  - Centrum Badan Klinicznych Pi-House, Poradnia Diabetologiczna, Gdansk, Pomeranian Voivodeship
  - Medica Pro Familia Sp. z o.o. Spolka Komandytowo Akcyjna, Oddzial w Gdyni, Gdynia, Pomeranian Voivodeship
  - Synexus Polska Sp. z o.o. Oddzial w Gdyni, Gdynia, Pomeranian Voivodeship
  - NZOZ "PRO CORDIS" Sopockie Centrum Badan Kardiologicznych, Gdynia, Pomeranian Voivodeship
  - Gabinet Kardiologiczno - lnternistyczny, Gdynia, Pomeranian Voivodeship
  - Centrum Medyczne "SOPMED" Sp. z o.o., Sopot, Pomeranian Voivodeship
  - Indywidualna Specjalistyczna Praktyka Lekarska Malgorzata Biedrzycka, Starogard Gdański, Pomeranian Voivodeship
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Wojewodzki Szpital Specjalistyczny Nr 4 w Bytomiu, Bytom, Silesian Voivodeship
  - Bogna Gabrylewicz Andrzej Ochala Unimed s.c., Katowice, Silesian Voivodeship
  - Pro Familia Altera Poradnia Wielospecjalistyczna, Katowice, Silesian Voivodeship
  - NZOZ Terapia Optima, Katowice, Silesian Voivodeship
  - Przychodnia Specjalistyczna Samodzielny Publiczny ZOZ w Rudzie Slaskiej,, Ruda Śląska, Silesian Voivodeship
  - NZOZ "Medyk"Sp. z o. o., Wola, Silesian Voivodeship
  - Wojewodzki Szpital Zespolony w Elblagu, Oddzial Kardiologiczny z Pododdzialem Kardiologii Inwazyjnej, Elblag, Warmian-Masurian Voivodeship
  - Specjalistyczny Osrodek Leczniczo-Badawczy Zbigniew Zegota, Ostróda, Warmian-Masurian Voivodeship
  - Centrum Medyczne AMED, Warsaw, WOJ Mazowieckie
  - Marek Piepiorka Gabinet Kardiologiczno - lnternistyczny, Gdynia
  - Nzoz Gall-Med, Krakow
  - NZOZ Centrum Zdrowia i Profilaktyki Dabie Sp. z.o.o., Krakow
  - "TWOJA PRZYCHODNIA" Sp. Z o.o, Lublin
  - Medicus w Opolu Sp z o. o., Opole
  - Centrum Zdrowia Metabolicznego Pawel Bogdanski, Poznan
  - NZOZ PRZYCHODNIA SPECJALISTYCZNA Andrzej Wittek Henryk Rudzki s.c., Ruda Śląska
  - KO-MED Centra Kliniczne Staszow, Staszów
  - Synexus Polska Sp. z o.o. Oddzial w Warszawie, Warsaw
  - Centrum Medyczne Warszawskiego Uniwersytetu Medycznego Sp. z o.o, Warsaw
  - Instytut Kardiologii im. Prymasa Tysiaclecia Stefana Kardynala Wyszynskiego Klinika Kardiologii, Warsaw
  - Synexus Polska Sp. z o.o. Oddzial we Wroclawiu, Wroclaw
  - Centrum Opieki Diabetologiczno-Endokrynologicznej i Ginekologiczno-Polozniczej, Wroclaw
  - Dobrostan Michal Bogacki, Wroclaw
  - Gabinet Lekarski Malgorzata Saryusz-Wolska, Lodz, Łódź Voivodeship
  - Specjalistyczny Osrodek Medycyny Wieku Dojrzalego Sp. z o.o. Jednostka 02, Lodz, Łódź Voivodeship
  - "Prywatny Gabinet Kardiologiczny" Dr N.Med. Maciej Kosmider, Lodz, Łódź Voivodeship
  - Niepubliczny Zaklad Opieki Zdrowotnej CEREO-MED Sp. z o.o., Lodz, Łódź Voivodeship
  - SPZOZ Centralny Szpital Kliniczny Uniwersytetu Medycznego w Lodzi 251 Pomorska, Lodz, Łódź Voivodeship
  - Prywatny Gabinet Lekarski Dr n. med. Michal Ogorek, Piotrkow Trybunalski, Łódź Voivodeship
  - Centrum Medyczne Ogrodowa Sp. z o.o., Skierniewice, Łódź Voivodeship
  - Prywatny Gabinet Lekarski Marianna Janion, Kielce, Świętokrzyskie Voivodeship
- Puerto Rico (8):
  - Endocrine Lipid Diabetes Research Institute, Ponce, PR
  - Miguel Sosa-Padilla, MD-Private Practice, San Juan, PR
  - Centro de Diabetes para Puerto Rico, San Juan, PR
  - The Office of Roberto J. Ayala-Rios, MD - Research Center and Private Practice (DMRA LLC), Añasco
  - Cardiometabolic Research Center, Inc., Ponce
  - Consultorio Medico Figueroa, San Juan
  - Pradnet Inc., San Juan
  - Altamira Family Medicine And Research Institute, San Juan
- Romania (30):
  - Pitesti-Arges County Emergency Hospital, Piteşti, Argeş
  - Medical Practice SRL, Oradea, Bihor County
  - County Clinical Emergency Hospital Oradea, Oradea, Bihor County
  - County Emergency Hospital Deva, Deva, Hunedoara County
  - Centrul Medical Sf. Stefan, Timișoara, JUD. Timis
  - Dr. Pop Calin Florin - Cabinet Cardiologie, Baia Mare, Maramureş
  - Podoleanu G. Cristian-Gheorghe-Calin - Cardiology Medical Practice, Târgu Mureş, Mureș County
  - Diabmed Dr. Popescu Alexandrina SRL, Diabet, Nutritie, Boli Metabolice, Ploieşti, Prahova
  - Dr. Busegeanu Mihaela Private Practice, Ploieşti, Prahova
  - Institute of Cardiovascular Diseases Timisoara, Timișoara, Timiș County
  - Euromedica Hospital, Baia Mare
  - S.C. Polimed Dacia S.R.L., Brasov
  - Centrul Medical de Diagnostic si Tratament Ambulator Neomed, Brasov
  - Spitalul Clinic Judetean De Urgenta Braila(Braila County Clincal Emergency Hospital), Brăila
  - Data Plus Medical Clinic, Bucharest
  - Spitalul Universitar De Urgenta Militar Central, Dr. Carol Davila, Bucharest
  - "Prof. Dr. N.C. Paulescu" National Institute of Diabetes, Nutrition and Metabolic Diseases,, Bucharest
  - Spitalul Clinic Colentina, Departament Cardiologie, Bucharest
  - SC Clinica Medicala Synexus SRL, Medicina Interna, Bucharest
  - SC Centrul Medical Policlinico Di Monza SRL, Cardiologie, Bucharest
  - SC Policlinica CCBR SRL, Bucharest
  - Med Plus SRL (Med Plus Ltd.), Bucharest
  - S.C. Centrul Medical "Sanatatea Ta" S.R.L., Bucharest
  - Spitalul Clinic Judetean de Urgenta Cluj-Napoca, Diabet Zaharat, Nutritie si Boli Metabolice, Cluj-Napoca
  - Dr. Mistodie Cristina Victoria MD, Office of, Galati
  - S.C. Diamed Obesity S.R.L., Galati
  - County Emergency Hospital Satu Mare Diabetes, Nutrition And Metabolic Diseases Department, Satu Mare
  - County Clinical Emergency Hospital Sibiu, Sibiu
  - Cardio Med SRL, Târgu Mureş
  - Centrul Medical Dr. Negrisanu SRL, Diabet Zaharat, Nutritie si Boli Metabolice, Timișoara
- Russia (72):
  - State Budgetary Healthcare Institution "Research Institution - Regional Clinical Hospital #1, Krasnodar, Krasnodarskiy Kray
  - State Budgetary Healthcare Institution Of Moscow Region "Lubertsy Regional Hospital #2", Lubertsy, Moscow Oblast
  - Federal State Budgetary Institution of Healthcare Hospital of Russian Academy of Sciences, Troitsk, Moscow Oblast
  - State Budgetary Institution "Ryazan Regional Clinical Hospital", Ryazan, Ryazan Oblast
  - Saint Petersburg State Budgetary Institution of Healthcare Municipal hospital, Saint Petersburg, Sestroretsk
  - FSBEI of HE Kazan State Medical University on the base of SBHI Clinical Hospital No.2, Kazan', Tatarstan Republic
  - SBEI of HPE Kazan State Medical University on the base of SBHI Clinical Hospital No.2, Kazan', Tatarstan Republic
  - Municipal Budgetary State Healthcare Institution "City Clinical Hospital #6", Chelyabinsk
  - Non-State Institution of Healthcare "Railway Clinical Hospital at station Chelyabinsk of open, Chelyabinsk
  - State Budgetary Healthcare Institution "Region Clinical Hospital #3", Chelyabinsk
  - Regional Budgetary Healthcare Institution "Cardiology Dispensary", Ivanovo
  - State Budgetary Institution of Healthcare of Kaluga Region "Kaluga Regional Hospital", Kaluga
  - Federal State Budgetary Educational Institution of Higher Education "Kazan State Medical University", Kazan'
  - State Autonomous Healthcare Institution, Kazan'
  - "SAHI of Kemerovo ""Regional Clinical Hospital of Emergency Medical Care n.a. M.A Podgorbunsky """, Kemerovo
  - Municipal Budgetary Institution of Healthcare, Kemerovo
  - Federal state budgetary institution Research institute of complex problems, Kemerovo
  - FSHI "Medical and Sanitary Unit of the Ministry of Internal Affairs of Russia across Kemerovo region, Kemerovo
  - Kirov Regional State Budgetary Healthcare Institution "Kirov City Clinical Hospital #1", Kirov
  - Regional Budgetary Healthcare Institution "Kursk City Clinical Emergency Hospital", Kursk
  - Non-State Institution of Healthcare "Central Clinical Hospital #6 OAO "RZhD", Moscow
  - Federal State Budgetary Institution "State Research Center for Preventive Medicine" of the Ministry, Moscow
  - SBHI of Moscow city "City Clinical Hospital #15 n.a. O.M. Filatova", Moscow
  - SBEI of HPE I. M. Sechenov First Moscow State Medical University, UKB #2, Moscow
  - State Healthcare Institution "City Clinical Hospital #51 of Healthcare Department of Moscow City", Moscow
  - Federal State Budgetary Institution "Central Clinical Hospital with Polyclinic", Moscow
  - Federal State Budgetary Institution "Russian Cardiology Research And Production Complex" Of Ministry, Moscow
  - Russian Cardiology Research And Production Complex of Ministry of Health of Russian Federation, Moscow
  - Moscow State Healthcare Institution "City clinical hospital n.a. S.P.Botkin", Moscow
  - SBIH "City Clinical Hospital #81 Departments of Healthcare of Moscow", Moscow
  - Federal State Budget Institution "Out-patient Clinic #3" of Russian Federation,, Moscow
  - State Regional Budgetary Healthcare Institution, Murmansk
  - State Budgetary Healthcare Institution of Nizhegorodskaya Region, Nizhny Novgorod
  - Federal State Budgetary Institution "Research Institute of Therapy and Preventive Medicine" of, Novosibirsk
  - SBRIHPE "Novosibirsk State Medical University" of MHSD of RF, Novosibirsk
  - "Reafan" LLC, Novosibirsk
  - "SBHI of Novosibirsk ""City Clinical Hospital of Emergency Medical Care # 2""", Novosibirsk
  - Municipal Budgetary Institution of Healthcare of Novosibirsk, Novosibirsk
  - State Budgetary Institution of Healthcare of Novosibirsk region City Clinical Hospital of Emergency, Novosibirsk
  - State Budgetary Institution of Healthcare"Penzenskaya Regional clinical hospital n.a N.N Burdenko", Penza
  - SBHI of Saint-Petersburg "City Hospital # 38 n.a. N.A. Semashko", Pushkin
  - Federal State Budgetary Educational Institution of Higher Education, Rostov-on-Don
  - State Budgetary Educational Institution Of Higher Professional Education, Rostov-on-Don
  - State Budgetary Educational Institution of Higher Professional Education, Rostov-on-Don
  - Limited Liability Company International Medical Centre SOGAZ, Saint Petersburg
  - Saint-Petersburg State Budgetary Institution of Healthcare "City Hospital #23", Saint Petersburg
  - Saint-Petersburg State Budgetary Healthcare Institution "City Alexandrovskaya Hospital", Saint Petersburg
  - Federal state budget institution of healthcare Saint-Petersburg clinical hospital of Russian Academy, Saint Petersburg
  - Limited Liability Company "Reavita", Saint Petersburg
  - "Limited Liability Company ""Institute of Medical Research""", Saint Petersburg
  - Limited Liability Company "Institute of Medical research", Saint Petersburg
  - LLC "Institution of medical studies", Saint Petersburg
  - City Hospital # 38 n.a. Semashko, Saint Petersburg
  - Federal State Budgetary Educational Institution of Higher Education, Saint Petersburg
  - SBEI of HPE "First Pavlov State Medical University of St. Petersburg" of the MOH of the RF, Saint Petersburg
  - Federal State Budgetary Institution "Advisory Diagnostic Center and Polyclinic", Saint Petersburg
  - Federal State Budgetary Institution, Saint Petersburg
  - Saint-Petersburg State Budgetary Healthcare Institution "City Hospital #15", Saint Petersburg
  - State Budgetary Healthcare Institution "Samara Regional Clinical Cardiology Dispensary", Samara
  - MHI "City Clinical Hospital #12" of the Healthcare Committee, Saratov
  - State Institution of Healthcare "Regional Clinical Hospital", Saratov
  - State Budget Educational Institution of Higher Professional Education, Smolensk
  - Tyumen Cardiology Research Center-branch of the Tomsk NRMC, Tomsk
  - GBOU VPO Siberian State Medical University Ministry of Healthcare of the Russian Federation, Tomsk
  - State Budgetary Educational Institution of Highest Professional Education "Siberian State Medical, Tomsk
  - State Autonomous Institution of Healthcare of the Tyumen region Tyumen Institute of Therapy, Tyumen
  - Affiliate of the Federal State Budgetary Institution Scientific Research Institute of Cardiology, Tyumen
  - State Autonomous Healthcare Institution of Yaroslavl region, Yaroslavl
  - FSBEI of HE "Yaroslavl State Medical University" MH of the Russian Federation, Yaroslavl
  - State Budgetary Healthcare Institution of Yaroslavl Region "Clinical Hospital No. 10", Yaroslavl
  - State Healthcare Institution of Yaroslavl Region "Clinical Hospital #8", Yaroslavl
  - Municipal Autonomous Institution "City Clinical Hospital #14", Yekaterinburg
- Slovakia (39):
  - Nemocnica Ruzinov-Univerzitna Nemocnica Bratislava (UNB), Bratislava, Bratislava Region
  - Stredoslovensky Ustav Srdcovych A Cievnych Chorob A.S., Banská Bystrica
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta Banska Bystrica, Banská Bystrica
  - Alian s.r.o., kardiologicka ambulancia, Bardejov
  - METABOL KLINIK s. r.o., Ambulancia pre diabetologiu, poruchy latkovej premeny a vyzivy, Bratislava
  - Univerzitna nemocnica Bratislava, Nemocnica Stare Mesto, l.intema klinika, Bratislava
  - Univerzitna nemocnica Bratislava, Nemocnica Stare Mesto, l.interna klinika, Bratislava
  - Univerzitna nemocnica Bratislava, Nemocnica Stare Mesto, Bratislava
  - UN Bratislava, Nemocnica Ruzinov, V. interna klinika LFUK a UN Bratislava, Bratislava
  - Kardiovaskularne centrum s.r.o., Bratislava
  - Metabolicke centrum MUDr. Katariny Raslovej, s.r.o., Bratislava
  - Narodny ustav srdcovych a cievnych chorob, a.s., Bratislava
  - Univerzitna Nemocnica Bratislava, Bratislava
  - KARDIO-SANUS spol., s.r.o., Bratislava
  - UN Bratislava Nemocnica Sv. Cyrila a Metoda, kardiologicka ambulancia 1, Bratislava
  - VERIA, s.r.o. -Kardiologicka ambulancia, Bratislava
  - Endiamed s.r.o. Nestatna diabetologicka a endokrinologicka ambulancia, Dolný Kubín
  - JM-Interna s.r.o., interna ambulancia, Dolný Kubín
  - CARDIO D&R s.r.o. , Kardiologicka ambulancia, Košice
  - AGTO., spol. s r. o., Košice
  - Cardio D&R spol.s.r.o., Kardiologicka ambulancia, Košice
  - Medicentrum Heart, Spol. S.R.O, Kráľovský Chlmec
  - CELL-B s.r.o. interna ambulancia, Levice
  - Liptovska nemocnica s poliklinikou MUDr.Ivana Stodolu Liptovsky Mikulas, Liptovský Mikuláš
  - KARDIO 1 s.r.o., Lučenec
  - Klinika hematologie a transfuziologie, Univerzitna nemocnica Martin, Martin
  - MEDI M&M s.r.o., Ambulancia vnutorneho lekarstva, Moldava nad Bodvou
  - MUDr. Kanderkova s.r.o., Diabetologicka ambulancia, Námestovo
  - Kardiocentrum Nitra s.r.o., kardiologicka ambulancia, Nitra
  - Fakultna Nemocnica s poliklinikou Nove Zamky, Nové Zámky
  - Mediab s.r.o. Diabetologicka ambulancia, Pezinok
  - BENIMED s.r.o., Piešťany
  - Medispol S.R.O., Prešov
  - Medilex s.r.o. Interna ambulancia, Rimavská Sobota
  - Kardioamb s.r.o., Rimavská Sobota
  - DIAMEL, s.r.o., Diabetologicka ambulancia, Trenčín
  - BV Medical, s.r.o. Diabetologicka ambulancia,, Trnava
  - Kardiologicka ambulancia, Trnava
  - Medivasa, s.r.o., Žilina
- South Africa (34):
  - Nash Ranjith Research Centre, Merebank, Durban
  - IATROS International, Bloemfontein, Free State
  - JOSHA Research, Bloemfontein, Free State
  - Welkom Clinical trial Centre, Welkom, Free State
  - Midrand Medical Centre, Halfway House, Gauteng
  - Sunward Park Hospital, Johannesburg, Gauteng
  - Sunninghill Hospital, Johannesburg, Gauteng
  - I Engelbrecht Research (Pty) Ltd, Lyttelton, Gauteng
  - Charlotte Maxeke Johannesburg Academic Hospital, Parktown, Gauteng
  - Medipark Centre for Clinical Research, Pretoria, Gauteng
  - Synexus Watermeyer Clinical Research Centre, Pretoria, Gauteng
  - Jongaie Research, Pretoria West, Gauteng
  - Roodepoort Medicross Clinical Research Centre, Roodepoort, Gauteng
  - Wits Clinical Research, Soweto, Gauteng
  - Medi-Clinic Heart Hospital, Sunnyside, Gauteng
  - Sunninghill Hospital, Sunninghill, Johannesburg
  - Glastonbury Medical Research Centre, Durban, KwaZulu-Natal
  - Suite 502, Durban, KwaZulu-Natal
  - Dr Ganesh c/o Dr NB Maharaj, Durban, KwaZulu-Natal
  - Limpopo Clinical Research Initiative, Thabazimbi, Limpopo
  - Zinakekele Medical centre, Moloto South, Mpumalanga
  - Drs Joynt Venter & Associates, Witbank (eMalahleni), Mpumalanga
  - Dr JM Engelbrecht Trial Site-Vergelegen Mediclinic, Cape Town, Western Cape
  - Tiervlei Trial Centre, Cape Town, Western Cape
  - Synopsis Research cc, Cape Town, Western Cape
  - Helderberg Research Institute, Somerset West, Western Cape
  - Synexus Helderberg Clinical Research Centre, Somerset West, Western Cape
  - Global Clinical Trials (Pty) Ltd., Arcadia, Pretoria
  - Unitas Hospital, Centurion
  - Clinresco Centres (Pty) Ltd-Central Professional Suits, Gauteng
  - Centre For Diabetes And Endocrinology, Johannesburg
  - Paarl Research Centre, Paarl
  - TREAD Research cc, Parow
  - Clinical Projects Research SA (Pty) Ltd, Worcester
- South Korea (21):
  - Chungbuk National University Hospital, Cheongju-si, Chungcheonbuk-do
  - Kangwon National University Hospital, Chuncheon, Gangwon-do
  - Yonsei University Wonju College of Medicine, Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Dongguk University Ilsan Hospital, Goyang-si, Gyeonggi-do
  - Inje University Ilsan Paik Hospital, Goyang-si, Gyeonggi-do
  - MyongJi Hospital, Goyang-si, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Uijeongbu St. Mary's Hospital-The Catholic University of Korea, Uijeongbu-si, Gyeonggi-do
  - Inha University Hospital, Jung-gu, Incheon
  - Hallym University Kangdong Sacred Heart Hospital, Seoul, Korea, Republic of
  - Inje University Busan Paik Hospital, Busan
  - Dong-A University Hospital, Busan
  - Daegu Catholic University Medical Center, Daegu
  - Konyang University Hospital, Daejeon
  - Daejeon St. Mary's Hospital-The Catholic University of Korea, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Gachon University Gil Medical Center, Incheon
  - Gangnam Severance Hospital, Yonsei University Health System, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - Asan Medical Center, Seoul
- Spain (77):
  - Hospital Clinico Universitario de Santiago de Compostela, Santiago de Compostela, A Coruna
  - Hospital Universitario de Santiago de Compostela, Santiago de Compostela, A Coruna
  - Hospital Virgen De Los Lirios, Alcoy, Alicante
  - Hospital General Comarcal de Elda Virgen de la Salud, Elda, Alicante
  - Hospital Regional Universitario de Malaga, Málaga, Andalusia
  - Hospital Universitario Virgen del Rocio, Seville, Andalusia
  - Hospital Comarcal d'Inca, Inca, Balearic Islands
  - Clinica Juaneda, Palma de Mallorca, Balearic Islands
  - Hospital Son Llatzer, Palma de Mallorca, Balearic Islands
  - Cap Florida, L'Hospitalet de Llobregat, Barcelona-cataluna
  - Hospital General de Granollers, Granollers, Barcelona/cataluña
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - CAP La Mina, Sant Adrià de Besòs, Barcelona
  - EAP Vic, Vic, Barcelona
  - Hospital Universitario de Cruces, Barakaldo, Basque Country
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Institut Catala De La Salut - Hospital Universitari Arnau De Vilanova (Huav), Lleida, Catalonia
  - Hospital Universitari de Tarragona Joan XXIII, Tarragona, Catalonia
  - Albera Salut, Peralada, Gerona
  - Hospital De Figueres, Figueres, Girona-catalonia
  - Hospital Arquitecto Marcide, Ferrol, LA Coruna
  - H. U. Principe de Asturias, Alcalá de Henares, Madrid
  - Hospital Principe de Asturias, Alcalá de Henares, Madrid
  - Hospital Universitario Principe de Asturias, Alcalá de Henares, Madrid
  - Hospital Universitario Fundacion Alcorcon, Alcorcón, Madrid
  - Hospital Universitario Puerta de Hierro - Majadahonda, Majadahonda, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Consultorio de Colloto, Colloto, Oviedo Asturias
  - Centro de Salud El Cristo, Oviedo, Principality of Asturias
  - Centro Salud Paulino Prieto, Oviedo, Principality of Asturias
  - Hospital Universitario Sant Joan de Reus, Reus, Tarragona
  - Hospital General de Requena, Requena, Valencia
  - Hospital Universitario San Juan de Alicante, San Juan de Alicante (Alicante), Valencia
  - Hospital Abente y Lago, A Coruña
  - Complejo Hospitalario Universitario A Coruna, A Coruña
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Hospital General Universitario de Alicante; Servicio Cardiologia, Alicante
  - Hospital Virgen del Mar, Almería
  - Parc de Salut mar ¿ Hospital del Mar, Barcelona
  - Parc De Salut Mar-Hospital Del Mar, Barcelona
  - Centre Teknon, Barcelona
  - EAP Sardenya, Barcelona
  - Hospital de la Santa Creu i Sant pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - CAP Centelles, Barcelona
  - Fundacio Hospital de I'Esperit Sant, Barcelona
  - Cap Disset De Setembre (Sant Cosme I Sant Damia), Barcelona/Cataluna
  - Hospital General De Granollers, Barcelona/Cataluña
  - H. General Universitario de Ciudad Real, Ciudad Real
  - Hospital Universitario Reina Sofia, Córdoba
  - Complexo Hospitalario Universitario Arquitecto Marcide-Profesor Novoa Santos De Ferrol, Ferrol
  - Hospital Universitario San Cecilio de Granada, Granada
  - Hospital Universitario Virgen de las Nieves (HUVN), Granada
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Universitario de La Princesa, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Carlos III, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario La Paz; Unidad Metabolico-Vascular, Madrid
  - Hospital Universitario Quiron Madrid, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Virgen De La Victoria, Málaga
  - Hospital General Universitario Morales Meseguer, Murcia
  - Clinica Nuevas Tecnologias en Diabetes y Endocrinologia, Seville
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario Virgen de Valme, Seville
  - CAP Muralles, Tarragona
  - Hospital General Universitario de Valencia, Valencia
  - Hospital Alvaro Cunqueiro (Hospital Meixoerio), Vigo
  - Hospital Clinico Universitario Miguel Servet; Medicina Interna, Zaragoza
- Sweden (23):
  - Karolinska Universitetssjukhuset Huddinge, Stockholm, Huddinge
  - Kasernens Läkarservice AB, Eksjö
  - Clinical Trial Center (CTC)/Centrum foer klinisk proevning, Gothenburg
  - Centrum for klinisk provning-Sahlgrenska Universitetssjukhus, Gothenburg
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Pharmasite AB, Helsingborg
  - Centralsjukhuset Karlstad, Karlstad
  - Centralsjukhuset Kristianstad, Kristianstad
  - Capio Citykliniken Hjartmottagning, Lund
  - Probar E Lund AB, Lund
  - Karlkliniken, Skanes Universitetssjukhus i Malmo, Malmo
  - Pharmasite, Malmo
  - Forskningsenheten, Medicinmottagningen Sahlgrenska Universitetssjukhuset/Molndal, Hus J, Mölndal
  - Ostersunds Sjukhus, Östersund
  - Dalecarlia Clinical Research Center, Rättvik
  - Skelleftea Lasarett, Skellefteå
  - Citydiabetes, Stockholm
  - Karolinska Trial Alliance, KTA Prim, Stockholm
  - Södersjukhuset Ab, Stockholm
  - Karolinska Universitetssjukhuset, Stockholm
  - Hjartkliniken, Stockholm
  - Akademiska Sjukhuset, Uppsala
  - Vastmanlands Sjukhus Vasteras, Västerås
- Switzerland (10):
  - Diagene Laboratories, Reinach, Basel Switzerland
  - Universitatsspital, Basel, Canton of Basel-City
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud
  - Policlinique Medicale Universitaire, Lausanne, Canton of Vaud
  - Kantonsspital Winterthur, Winterthur, Canton of Zurich
  - Fondazione Diabete Lugano, Lugano, Canton Ticino
  - Hopitaux Universitaires de Geneve, Geneva
  - Luzerner Kantonsspital Luzern, Lucerne
  - Cardiocentro Ticino, Lugano
  - Kantonsspital St. Gallen, Sankt Gallen
- Taiwan (8):
  - China Medical University Hospital, Taichung, Taiwan R O C
  - Chung Shan Medical University Hospital, Taichung, Taiwan ROC
  - Kaohsiung Medical University Chung-Ho Memorial Hospital - New, Kaohsiung City
  - National Cheng Kung University (NCKU) Hospital, Tainan
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - MacKay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Thailand (8):
  - Division of Cardiology, Department of Medicine, Faculty of Medicine, Siriraj Hospital, Mahidol, Bangkoknoi, Bangkok
  - Clinical Research Center, Phramongkutklao Hospital, Rajathevee, Bangkok
  - Endocrine Unit, Department of Medicine, Phramongkutklao Hospital, Rajathevee, Bangkok
  - Cardiology Unit, Department of Medicine, Faculty of Medicine,Ramathibodi Hospital,Mahidol University, Ratchathewi, Bangkok
  - Division of Cardiology, Department of medicine,Faculty of Medicine, Srinagarind Hospital, Khon Kaen, Muang, Changwat Khon Kaen
  - Division of Cardiology, Department of Medicine, Faculty of Medicine, Songklanagarind Hospital,, Hat Yai, Changwat Songkhla
  - Heart Center, Songklanagarind Prince of Songkla University, Hat Yai, Changwat Songkhla
  - Division Of cardiology,Department of Medicine,Faculty Of Medicine,Chulalongkorn University, Bangkok
- Turkey (Türkiye) (20):
  - Dokuz Eylul Univesitesi Tip Fakultesi Hastanesi, Izmir, Ankara
  - Baskent University, Adana Yuregir Training & Research Hospital, Adana
  - A.karahisar Kocatepe Universitesi Hastanesi Ahmet Necdet Sezer Uygulama ve Arastirma Hastanesi, Afyonkarahisar
  - Diskapi Yildirim Beyazit Egitim ve Arastirma Hastanesi, Ankara
  - Akdeniz Universitesi Tip Fakultesi Hastanesi, Antalya
  - Akdeniz Universitesi Tip Fakultesi, Antalya
  - Antalya Training & Research Hospital, Antalya
  - Bursa Yuksek Ihtisas Egitim ve Arastirma Hastanesi, Bursa
  - Gaziantep Universitesi Tip Fakultesi Sahinbey Egitim ve Arastirma Hastanesi, Gaziantep
  - Bezmialem Vakif Universitesi Tip Fakultesi Kardiyoloji Anabilim Dali, Istanbul
  - Bezmialem Vakif Universitesi Tip Fakultesi Kardiyoloji Bolumu, Istanbul
  - Istanbul Universitesi Istanbul Tip Fakultesi, Istanbul
  - Istanbul Universitesi Kardiyoloji Enstitusu, Istanbul
  - Yeditepe University School of Medicine, Istanbul
  - Ege University, School of Medicine, Izmir
  - Dokuz Eylul Universitesi Tip Fakultesi, Izmir
  - Kocaeli University School Of Medicine-Kocaeli Universitesi Tip Fakultesi, Kocaeli
  - Dumlupinar Universitesi Kutahya Evliya Celebi EAH, Kütahya
  - Mersin University, School of Medicine, Mersin
  - Recep Tayyip Erdogan University School of Medicine, Training & Research Hospital, Rize
- United Kingdom (56):
  - Synexus Thames Valley Clinical Research Centre, Reading, Berkshire
  - Westongrove Research Centre, Aylesbury, Buckinghamshire
  - Peterborough City Hospital, Peterborough, Cambridgeshire
  - Morrab Surgery, Penzance, Cornwall
  - Brannel Surgery, St Austell, Cornwall
  - The Michael White Centre for Diabetes & Endocrinology, Hull Royal Infirmary, Hull, EAST Yorkshire
  - Queen's Hospital, Romford, Essex
  - Synexus Manchester Clinical Research Centre-Manchester Science Park, Manchester, Greater Manchester
  - Royal Oldham Hospital, Oldham, Greater Manchester
  - St Francis Surgery, Chandlers Ford, Hampshire
  - Lister Hospital, Stevenage, Hertfordshire
  - East and North Hertfordshire NHS Trust, Welwyn Garden City, Hertfordshire
  - Howlands Clinic - Queen Elizabeth II Hospital, Welwyn Garden City, Hertfordshire
  - Synexus Scotland Clinical Research Centre, Glasgow, Lanarkshire
  - Layton Medical Centre, Blackpool, Lancashire
  - Synexus Lancashire Clinical Research Centre, Chorley, Lancashire
  - Salford Royal NHS Foundation Trust - Dermatology Centre, Salford, M6 8HD
  - Synexus Merseyside Clinical Research Centre, Liverpool, Merseyside
  - The Royal Liverpool and Broadgreen -University Hospitals NHS Trust, Liverpool, Merseyside
  - Whitby Group Practice, Whitby, North Yorkshire
  - Albany House Medical Centre, Wellingborough, Northants
  - Southern Health & Social Care Trust, Craigavon Area Hospital, Portadown, Northern Ireland
  - Synexus North East Clinical Research Centre - Hexham General Hospital, Hexham, Northumberland
  - South Axholme Practice, Doncaster, South Yorkshire
  - Central Manchester University Hospitals NHS Foundation Trust, Manchester, South Yorkshire
  - The Crouch Oak Family Practice, Addlestone, Surrey
  - Ely Bridge Surgery, Cardiff, Wales
  - Synexus Midlands Clinical Research Centre, Birmingham, WEST Midlands
  - City Hospital, Birmingham, WEST Midlands
  - Heart of England NHS Trust, Birmingham, WEST MIDS
  - Prince Philip Hospital, Llanelli, WEST Wales
  - Royal Free London NHS Foundation Trust, Barnet
  - Royal Victoria Hospital, Belfast
  - Laurie Pike Health Centre, Birmingham
  - Heart of England NHS Foundation Trust, Dept. of Clinical Biochemistry & Immunology, Birmingham
  - Royal Bolton Hospital - Bolton Nhs Foundation Trust, Bolton
  - Synexus Wales Clinical Research Centre, Cardiff
  - Ashgate Medical Practice, Chesterfield
  - Conquest Hospital - East Sussex Healthcare NHS Trust, East Sussex
  - Little Common Surgery, East Sussex
  - Sea Road Surgery, East Sussex
  - Staploe Medical Centre, Ely
  - The Queen Elizabeth University Hospital- NHS Greater Glasgow and Clyde, Glasgow
  - McGlone Practice Baillieston Health Centre, Glasgow
  - Burbage Surgery, Hinckley
  - William Harvey Heart Centre (WHHC), London
  - Royal Free Hospital, London
  - Peart-Rose Research Unit, Hammersmith Hospital, Imperial College NHS Trust, London
  - The Red Porto cabin, The James Cook University Hospital, Middlesbrough
  - St Mary's Hospital, Newport
  - Wansford And Kings Cliffe Practice, Peterborough
  - Rothwell and Desborough Healthcare Group, Rothwell, Northants
  - Abertawe Bro Morgannwg University Local Health Board, Swansea
  - Western Sussex Hospitals NHS Trust, Worthing
  - York Medical Group, York
  - Strensall Healthcare Centre, York

REFERENCES:
- [Derived] Chasman DI, Hyde CL, Giulianini F, Danning RD, Wang EQ, Hickling T, Ridker PM, Loomis AK. Genome-wide pharmacogenetics of anti-drug antibody response to bococizumab highlights key residues in HLA DRB1 and DQB1. Sci Rep. 2022 Mar 11;12(1):4266. doi: 10.1038/s41598-022-07997-5. PMID 35277540
- [Derived] Pradhan AD, Aday AW, Rose LM, Ridker PM. Residual Inflammatory Risk on Treatment With PCSK9 Inhibition and Statin Therapy. Circulation. 2018 Jul 10;138(2):141-149. doi: 10.1161/CIRCULATIONAHA.118.034645. Epub 2018 May 1. PMID 29716940
- [Derived] Ridker PM, Rose LM, Kastelein JJP, Santos RD, Wei C, Revkin J, Yunis C, Tardif JC, Shear CL; Studies of PCSK9 Inhibition and the Reduction of vascular Events (SPIRE) Investigators. Cardiovascular event reduction with PCSK9 inhibition among 1578 patients with familial hypercholesterolemia: Results from the SPIRE randomized trials of bococizumab. J Clin Lipidol. 2018 Jul-Aug;12(4):958-965. doi: 10.1016/j.jacl.2018.03.088. Epub 2018 Apr 3. PMID 29685591
- [Derived] Ridker PM, Revkin J, Amarenco P, Brunell R, Curto M, Civeira F, Flather M, Glynn RJ, Gregoire J, Jukema JW, Karpov Y, Kastelein JJP, Koenig W, Lorenzatti A, Manga P, Masiukiewicz U, Miller M, Mosterd A, Murin J, Nicolau JC, Nissen S, Ponikowski P, Santos RD, Schwartz PF, Soran H, White H, Wright RS, Vrablik M, Yunis C, Shear CL, Tardif JC; SPIRE Cardiovascular Outcome Investigators. Cardiovascular Efficacy and Safety of Bococizumab in High-Risk Patients. N Engl J Med. 2017 Apr 20;376(16):1527-1539. doi: 10.1056/NEJMoa1701488. Epub 2017 Mar 17. PMID 28304242
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1481022&StudyName=The%20Evaluation%20Of%20PF-04950615%20%28RN316%29%2C%20In%20Reducing%20The%20Occurrence%20Of%20Major%20Cardiovascular%20Events%20In%20High%20Risk%20Subjects

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received single dose of placebo matched to PF-04950615 subcutaneous injection once every 2 weeks for upto 3 years. Participants were followed up to 40 days after the last dose.
- Bococizumab (PF-04950615): Participants received single dose of PF-04950615 150 milligrams, subcutaneous injection once every 2 weeks for upto 3 years. Participants were followed up to 40 days after the last dose.
Period: Overall Study
Arm/Group | Placebo | Bococizumab (PF-04950615)
Started | 8390 | 8394
Treated | 8374 | 8386
Completed | 8164 | 8177
Not Completed | 226 | 217
Not completed — Adverse Event | 5 | 5
Not completed — Death | 65 | 72
Not completed — Lost to Follow-up | 70 | 66
Not completed — Withdrew consent | 68 | 62
Not completed — Other | 2 | 4
Not completed — Randomized, Not Treated | 16 | 8

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): all participants who were randomized, excluding who attempted to be randomized more than once into a bococizumab cardiovascular (CV) outcomes trial (B1481022/B1481038) or attempted to be randomized in more than 1 CV outcomes trial and all participants enrolled at study Site 3027 where a quality-related event was identified.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Bococizumab (PF-04950615) | Total
Number analyzed (Participants) | 8390 | 8394 | 16784
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.3 (9.2) | 63.3 (9.1) | 63.3 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2223 | 2207 | 4430
  Male | 6167 | 6187 | 12354
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1758 | 1746 | 3504
  Not Hispanic or Latino | 6631 | 6642 | 13273
  Unknown or Not Reported | 1 | 6 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 354 | 369 | 723
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 392 | 412 | 804
  White | 7315 | 7280 | 14595
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 329 | 333 | 662

OUTCOME MEASURES:

1. Primary Outcome: Event Rate Per 100 Participant-Years For First Occurrence of Major Cardiovascular (CV) Event
Description: Event rate per 100 participant-years for first occurrence of major CV event (adjudicated by Adjudication Committee) was reported. Major CV event was defined as any of the following: CV death (defined as sudden cardiac death, fatal myocardial infarction [MI], death due to heart failure, death due to stroke [fatal ischemic stroke or fatal stroke of undetermined etiology], or death due to other cardiovascular causes) non-fatal MI, non-fatal stroke, and hospitalization for unstable angina needing urgent revascularization. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of major CV event (maximum duration: up to 3.4 years)
Population: Full analysis set (FAS): all participants who were randomized, excluding who attempted to be randomized more than once into a bococizumab CV outcomes trial (B1481022/B1481038) or attempted to be randomized in more than 1 CV outcomes trial and all participants enrolled at study Site 3027 where a quality-related event was identified.
Measure: Number (95% Confidence Interval); unit: Events Per 100 Participant-Years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 8390 | 8394
Events Per 100 Participant-Years | 3.02 [2.59 to 3.51] | 3.01 [2.58 to 3.50]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); Hazard ratio and 95 percent (%) Confidence Interval (CI) were from a Cox proportional hazards model stratified by geographic region and low density lipoprotein cholesterol (LDL-C) at pre-screening (less than [<] 100 milligrams per deciliters [mg/dL], greater than and equal to [>=] 100 mg/dL) with treatment as a co-variate; Test type: Superiority; p = 0.930905, Log Rank; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.80 to 1.22]

2. Secondary Outcome: Event Rate Per 100 Participant-Years For First Occurrence of Composite Endpoint of Cardiovascular Death, Non-Fatal Myocardial Infraction, or Non-Fatal Stroke
Description: Event rate per 100 participant-years for first occurrence of composite endpoint of CV death, non-fatal MI or non-fatal stroke (adjudicated by Adjudication Committee) was reported. Cardiovascular death was defined as sudden cardiac death, fatal MI, death due to heart failure, death due to stroke (fatal ischemic stroke or fatal stroke of undetermined etiology), or death due to other cardiovascular causes. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of the CV death, non-fatal MI or non-fatal stroke (maximum duration: up to 3.4 years)
Population: FAS: all participants who were randomized, excluding who attempted to be randomized more than once into a bococizumab CV outcomes trial (B1481022/B1481038) or attempted to be randomized in more than 1 CV outcomes trial and all participants enrolled at study Site 3027 where a quality-related event was identified.
Measure: Number (95% Confidence Interval); unit: Events Per 100 Participant-Years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 8390 | 8394
Events Per 100 Participant-Years | 2.49 [2.10 to 2.93] | 2.59 [2.19 to 3.04]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); Hazard ratio and 95% CI were from a Cox proportional hazards model stratified by geographic region and LDL-C at pre-screening (<100 mg/dL, >=100 mg/dL) with treatment as a covariate; Test type: Superiority; p = 0.784265, Log Rank; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.82 to 1.30]

3. Secondary Outcome: Event Rate Per 100 Participant-Years For First Occurrence of Composite Endpoint of All-Cause Death, Non-Fatal Myocardial Infraction, Non-Fatal Stroke, or Hospitalization for Unstable Angina Needing Urgent Revascularization
Description: Event rate per 100 participant-years for first occurrence of composite endpoint of all-cause death, non-fatal MI, non-fatal stroke, or hospitalization for unstable angina needing urgent revascularization (adjudicated by Adjudication Committee) was reported. All-cause death was defined as the death due to any cause during the course of study. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of all-cause death, non-fatal MI, non-fatal stroke, or hospitalization for unstable angina needing urgent revascularization (maximum duration: up to 3.4 years)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events Per 100 Participant-Years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 8390 | 8394
Events Per 100 Participant-Years | 3.51 [3.04 to 4.03] | 3.48 [3.02 to 4.00]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.892441, Log Rank; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.81 to 1.20]

4. Secondary Outcome: Event Rate Per 100 Participant-Years For First Occurrence of Composite Endpoint of All-Cause Death, Non-Fatal Myocardial Infarction, or Non-Fatal Stroke
Description: Event rate per 100 participant-years for first occurrence of composite endpoint of all-cause death, non-fatal MI, or non-fatal stroke (adjudicated by adjudication committee) was reported. All-cause death was defined as the death due to any cause during the course of study. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of the all-cause death, non-fatal MI, or non-fatal stroke (maximum duration: up to 3.4 years)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events Per 100 Participant-Years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 8390 | 8394
Events Per 100 Participant-Years | 2.98 [2.55 to 3.46] | 3.06 [2.62 to 3.54]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.845797, Log Rank; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.83 to 1.26]

5. Secondary Outcome: Event Rate Per 100 Participant-Years For First Occurrence of Hospitalization for Unstable Angina Needing Urgent Revascularization
Description: Event rate per 100 participant-years for first occurrence of hospitalization for unstable angina needing urgent revascularization (adjudicated by adjudication committee) was reported. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of hospitalization for unstable angina needing urgent revascularization (maximum duration: up to 3.4 years)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events Per 100 Participant-Years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 8390 | 8394
Events Per 100 Participant-Years | 0.57 [0.39 to 0.80] | 0.47 [0.31 to 0.68]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.431903, Log Rank; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.49 to 1.36]

6. Secondary Outcome: Event Rate Per 100 Participant-Years For First Occurrence of Composite Endpoint of Cardiovascular Death, Non-Fatal Myocardial Infarction, Non-Fatal Stroke and Hospitalization for Unstable Angina
Description: Event rate per 100 participant-years for first occurrence of composite endpoint of cardiovascular death, non-fatal MI, non-fatal stroke and hospitalization for unstable angina (adjudicated by adjudication committee) was reported. Cardiovascular death was defined as sudden cardiac death, fatal MI, death due to heart failure, death due to stroke (fatal ischemic stroke or fatal stroke of undetermined etiology), or death due to other cardiovascular causes. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of cardiovascular death, non-fatal MI, non-fatal stroke and hospitalization for unstable angina (maximum duration: up to 3.4 years)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events Per 100 Participant-Years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 8390 | 8394
Events Per 100 Participant-Years | 3.22 [2.77 to 3.72] | 3.19 [2.74 to 3.69]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.883797, Log Rank; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.80 to 1.21]

7. Secondary Outcome: Event Rate Per 100 Participant-Years For Cardiovascular Death
Description: Event rate per 100 participant-years for cardiovascular death (adjudicated by adjudication committee) was reported. Cardiovascular death was defined as sudden cardiac death, fatal MI, death due to heart failure, death due to stroke (fatal ischemic stroke or fatal stroke of undetermined etiology), or death due to other cardiovascular causes. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of adjudicated and confirmed occurrence of cardiovascular death (maximum duration: up to 3.4 years)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events Per 100 Participant-Years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 8390 | 8394
Events Per 100 Participant-Years | 0.52 [0.35 to 0.74] | 0.64 [0.45 to 0.88]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.455690, Log Rank; Hazard Ratio (HR) = 1.20, 95% CI 2-sided [0.74 to 1.95]

8. Secondary Outcome: Event Rate Per 100 Participant-Years For First Occurrence of Any Myocardial Infarction (Fatal or Non-Fatal)
Description: Event rate per 100 participant-years for first occurrence of any MI (fatal or non-fatal) (adjudicated by adjudication committee) was reported. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of any MI (fatal or non-fatal) (maximum duration: up to 3.4 years)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events Per 100 Participant-Years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 8390 | 8394
Events Per 100 Participant-Years | 1.56 [1.26 to 1.92] | 1.74 [1.41 to 2.11]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.469496, Log Rank; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.84 to 1.48]

9. Secondary Outcome: Event Rate Per 100 Participant-Years For Fatal Myocardial Infarction
Description: Event rate per 100 participant-years for fatal MI (adjudicated by adjudication committee) was reported. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of adjudicated and confirmed occurrence of fatal MI (maximum duration: up to 3.4 years)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events Per 100 Participant-Years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 8390 | 8394
Events Per 100 Participant-Years | 0.03 [0.00 to 0.12] | 0.05 [0.01 to 0.15]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.633022, Log Rank; Hazard Ratio (HR) = 1.54, 95% CI 2-sided [0.26 to 9.23]

10. Secondary Outcome: Event Rate Per 100 Participant-Years For First Occurrence of Non-Fatal Myocardial Infarction
Description: Event rate per 100 participant-years for first occurrence of non-fatal MI (adjudicated by adjudication committee) was reported. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of non-fatal MI (maximum duration: up to 3.4 years)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events Per 100 Participant-Years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 8390 | 8394
Events Per 100 Participant-Years | 1.53 [1.23 to 1.88] | 1.70 [1.38 to 2.07]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.467650, Log Rank; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.83 to 1.48]

11. Secondary Outcome: Event Rate Per 100 Participant-Years For First Occurrence of Any Stroke (Fatal or Non-Fatal)
Description: Event rate per 100 participant-years for first occurrence of any stroke (fatal or non-fatal) (adjudicated by adjudication committee) was reported. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of any stroke (fatal or non-fatal) (maximum duration: up to 3.4 years)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events Per 100 Participant-Years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 8390 | 8394
Events Per 100 Participant-Years | 0.71 [0.51 to 0.96] | 0.38 [0.24 to 0.57]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.015462, Log Rank; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.32 to 0.89]

12. Secondary Outcome: Event Rate Per 100 Participant-Years For First Occurrence of Any Stroke (Fatal or Non-Fatal), of Any Etiology
Description: Event rate per 100 participant-years for first occurrence of any stroke (fatal or non-fatal), of any etiology (adjudicated by adjudication committee) was reported. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of any stroke (fatal or non-fatal), of any etiology (maximum duration: up to 3.4 years)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events Per 100 Participant-Years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 8390 | 8394
Events Per 100 Participant-Years | 0.79 [0.58 to 1.06] | 0.43 [0.28 to 0.64]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.011863, Log Rank; Hazard Ratio (HR) = 0.54, 95% CI 2-sided [0.33 to 0.88]

13. Secondary Outcome: Event Rate Per 100 Participant-Years For Fatal Stroke
Description: Event rate per 100 participant-years for fatal stroke (adjudicated by adjudication committee) was reported. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of fatal stroke (maximum duration: up to 3.4 years)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events Per 100 Participant-Years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 8390 | 8394
Events Per 100 Participant-Years | 0.10 [0.04 to 0.22] | 0.05 [0.01 to 0.15]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.316066, Log Rank; Hazard Ratio (HR) = 0.50, 95% CI 2-sided [0.12 to 2.00]

14. Secondary Outcome: Event Rate Per 100 Participant-Years For First Occurrence of Non-Fatal Stroke
Description: Event rate per 100 participant-years for first occurrence of non-fatal stroke (adjudicated by adjudication committee) was reported. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of non-fatal stroke (maximum duration: up to 3.4 years)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events Per 100 Participant-Years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 8390 | 8394
Events Per 100 Participant-Years | 0.62 [0.44 to 0.86] | 0.33 [0.20 to 0.51]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.020328, Log Rank; Hazard Ratio (HR) = 0.52, 95% CI 2-sided [0.30 to 0.91]

15. Secondary Outcome: Event Rate Per 100 Participant-Years For First Occurrence of Hospitalization for Unstable Angina
Description: Event rate per 100 participant-years for first occurrence of hospitalization for unstable angina (adjudicated by adjudication committee) was reported. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of hospitalization for unstable angina (maximum duration: up to 3.4 years)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events Per 100 Participant-Years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 8390 | 8394
Events Per 100 Participant-Years | 0.78 [0.57 to 1.04] | 0.64 [0.45 to 0.88]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.367069, Log Rank; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.53 to 1.27]

16. Secondary Outcome: Event Rate Per 100 Participant-Years For First Occurrence of Hospitalization for Congestive Heart Failure (CHF)
Description: Event rate per 100 participant-years for first occurrence of hospitalization for CHF (adjudicated by adjudication committee) was reported. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of hospitalization for congestive heart failure (maximum duration: up to 3.4 years)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events Per 100 Participant-Years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 8390 | 8394
Events Per 100 Participant-Years | 0.81 [0.60 to 1.08] | 0.69 [0.49 to 0.94]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.443081, Log Rank; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.56 to 1.29]

17. Secondary Outcome: Event Rate Per 100 Participant-Years For First Occurrence of Coronary Revascularization
Description: Event rate per 100 participant-years for first occurrence of coronary revascularization (adjudicated by adjudication committee) was reported. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of coronary revascularization (maximum duration: up to 3.4 years)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events Per 100 Participant-Years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 8390 | 8394
Events Per 100 Participant-Years | 2.74 [2.33 to 3.20] | 2.45 [2.06 to 2.89]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.343817, Log Rank; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.71 to 1.12]

18. Secondary Outcome: Event Rate Per 100 Participant-Years For First Occurrence of Coronary Artery Bypass Graft Surgery (CABG)
Description: Event rate per 100 participant-years for first occurrence of CABG (adjudicated by adjudication committee) was reported. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of CABG (maximum duration: up to 3.4 years)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events Per 100 Participant-Years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 8390 | 8394
Events Per 100 Participant-Years | 0.40 [0.25 to 0.60] | 0.41 [0.26 to 0.61]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.889065, Log Rank; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.59 to 1.85]

19. Secondary Outcome: Event Rate Per 100 Participant-Years For First Occurrence of Percutaneous Coronary Intervention (PCI)
Description: Event rate per 100 participant-years for first occurrence of PCI (adjudicated by adjudication committee) was reported. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of PCI (maximum duration: up to 3.4 years)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events Per 100 Participant-Years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 8390 | 8394
Events Per 100 Participant-Years | 2.37 [1.99 to 2.80] | 2.08 [1.73 to 2.49]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.308388, Log Rank; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.69 to 1.13]

20. Secondary Outcome: Event Rate Per 100 Participant-Years For First Occurrence of Any Arterial Revascularizations
Description: Event rate per 100 participant-years for first occurrence of any arterial revascularizations (adjudicated by adjudication committee) was reported. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of first adjudicated and confirmed occurrence of any arterial revascularizations (maximum duration: up to 3.4 years)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events Per 100 Participant-Years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 8390 | 8394
Events Per 100 Participant-Years | 1.26 [0.99 to 1.59] | 1.28 [1.00 to 1.61]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.874835, Log Rank; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.74 to 1.42]

21. Secondary Outcome: Event Rate Per 100 Participant-Years For All-Cause Death
Description: Event rate per 100 participant-years for all-cause death (adjudicated by adjudication committee) was reported. All-cause death was defined as the death due to any cause during the course of study. Event rate was calculated as the number of events per 100 participant-years at risk.
Time Frame: From baseline until the date of adjudicated and confirmed occurrence of all-cause death (maximum duration: up to 3.4 years)
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events Per 100 Participant-Years
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 8390 | 8394
Events Per 100 Participant-Years | 1.00 [0.76 to 1.29] | 1.13 [0.88 to 1.44]
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.526269, Log Rank; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.79 to 1.60]

22. Secondary Outcome: Percent Change From Baseline in Low Density Lipoprotein Cholesterol at Week 14
Time Frame: Baseline, Week 14
Population: Analysis was performed on FAS. Here, "Number of participants analyzed "(N) signifies those participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 6448 | 6439
Percent change | 3.40 (0.31) | -57.17 (0.31)
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); Lease Square (LS)- mean differences, associated 95% CI, and p-values were from a mixed model repeated measures (MMRM) model including observations through Week 70 with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographic region and LDL-C at pre-screening (<100 mg/dL, >=100 mg/dL); Test type: Superiority; p < 0.001, Mixed Effect Model Repeat Measurement; LS-mean difference = -60.57, 95% CI 2-sided [-61.43 to -59.71]

23. Secondary Outcome: Nominal Change From Baseline in Low Density Lipoprotein Cholesterol at Week 14
Time Frame: Baseline, Week 14
Population: Analysis was performed on FAS. Here, "N" signifies number of participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 6448 | 6439
mg/dL | 2.33 (0.28) | -52.37 (0.28)
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); LS- mean differences and associated 95% CI, and p-values were from an MMRM model including observations through Week 70 with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographic region and LDL-C at pre-screening (<100 mg/dL, >=100 mg/dL); Test type: Superiority; p < 0.001, Mixed Effect Model Repeat Measurement; LS-mean difference = -54.70, 95% CI 2-sided [-55.48 to -53.92]

24. Secondary Outcome: Percent Change From Baseline in Low Density Lipoprotein Cholesterol at Last Post-Baseline Measurement
Time Frame: Baseline, last post-baseline measurement (any time up to Week 140)
Population: Analysis was performed on FAS. Here, "N" signifies number of participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 8240 | 8254
Percent Change | 5.05 (0.35) | -41.67 (0.35)
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); LS- mean difference and associated 95% CI, and p-value were from an analysis of covariance (ANCOVA) model with fixed effects for treatment group, baseline value, geographic region and LDL-C at pre-screening (<100 mg/dL, >=100 mg/dL); Test type: Superiority; p < 0.001, ANCOVA; LS-mean difference = -46.72, 95% CI 2-sided [-47.68 to -45.76]

25. Secondary Outcome: Percent Change From Baseline in Lipid Levels at Week 14
Description: Lipids included non-high density lipoprotein cholesterol (non-HDL-C), total cholesterol, very low density lipoprotein cholesterol (VLDL-C), remnant lipoprotein cholesterol (RLP-C), apolipoprotein B (Apo B), HDL-C and apolipoprotein A-I (Apo A-I).
Time Frame: Baseline, Week 14
Population: Analysis was performed on FAS. Here, number analyzed "n" signifies number of participants who were evaluable for the specified categories.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 8390 | 8394
Percent Change
  Non - HDL-C: number analyzed (Participants) | 6427 | 6412
  Non - HDL-C | 3.21 (0.28) | -51.66 (0.28)
  Total cholesterol: number analyzed (Participants) | 6441 | 6431
  Total cholesterol | 2.38 (0.20) | -34.13 (0.20)
  VLDL - C: number analyzed (Participants) | 6443 | 6433
  VLDL - C | 6.52 (0.45) | -13.65 (0.45)
  RLP - C: number analyzed (Participants) | 6418 | 6400
  RLP - C | 9.23 (0.79) | -21.02 (0.79)
  Apo B: number analyzed (Participants) | 5887 | 5894
  Apo B | 2.80 (0.31) | -55.76 (0.31)
  HDL - C: number analyzed (Participants) | 6431 | 6412
  HDL - C | 1.19 (0.16) | 7.33 (0.16)
  Apo A - I: number analyzed (Participants) | 5890 | 5896
  Apo A - I | 1.21 (0.18) | 4.74 (0.18)
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); Non-HDL-C: LS- mean differences, associated 95% CI, and p-values were from an MMRM model including observations through Week 70 with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographic region and LDL-C at pre-screening (<100 mg/dL, >=100 mg/dL); Test type: Superiority; p < 0.001, Mixed Effect Model Repeat Measurement; LS-mean difference = -54.88, 95% CI 2-sided [-55.66 to -54.09]
Statistical Analysis 2: Comparison: Placebo vs Bococizumab (PF-04950615); Total cholesterol: LS- mean differences, associated 95% CI, and p-values were from an MMRM model including observations through Week 70 with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographic region and LDL-C at pre-screening (<100 mg/dL, >=100 mg/dL); Test type: Superiority; p < 0.001, Mixed Effect Model Repeat Measurement; LS-mean difference = -36.51, 95% CI 2-sided [-37.07 to -35.95]
Statistical Analysis 3: Comparison: Placebo vs Bococizumab (PF-04950615); VLDL-C: LS- mean differences, associated 95% CI, and p-values were from an MMRM model including observations through Week 70 with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographic region and LDL-C at pre-screening (<100 mg/dL, >=100 mg/dL); Test type: Superiority; p < 0.001, Mixed Effect Model Repeat Measurement; LS-mean difference = -20.17, 95% CI 2-sided [-21.42 to -18.93]
Statistical Analysis 4: Comparison: Placebo vs Bococizumab (PF-04950615); RLP-C: LS- mean differences, associated 95% CI, and p-values were from an MMRM model including observations through Week 70 with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographic region and LDL-C at pre-screening (<100 mg/dL, >=100 mg/dL); Test type: Superiority; p < 0.001, Mixed Effect Model Repeat Measurement; LS-Mean Difference = -30.25, 95% CI 2-sided [-32.44 to -28.07]
Statistical Analysis 5: Comparison: Placebo vs Bococizumab (PF-04950615); Apo B: LS -mean differences, associated 95% CI, and p-values were from an MMRM model including observations through Week 52 with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographic region and LDL-C at pre-screening (<100 mg/dL, >=100 mg/dL); Test type: Superiority; p < 0.001, Mixed Effect Model Repeat Measurement; LS-Mean Difference = -58.55, 95% CI 2-sided [-59.42 to -57.69]
Statistical Analysis 6: Comparison: Placebo vs Bococizumab (PF-04950615); HDL-C: LS- mean differences, associated 95% CI, and p-values were from an MMRM model including observations through Week 70 with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographic region and LDL-C at pre-screening (<100 mg/dL, >=100 mg/dL); Test type: Superiority; p < 0.001, Mixed Effect Model Repeat Measurement; LS-Mean Difference = 6.14, 95% CI 2-sided [5.69 to 6.59]
Statistical Analysis 7: Comparison: Placebo vs Bococizumab (PF-04950615); Apo A-I: LS- mean differences, associated 95% CI, and p-values were from an MMRM model including observations through Week 52 with fixed effects for treatment group, visit, treatment group*visit interaction, baseline value, baseline value*visit interaction, geographic region and LDL-C at pre-screening (<100 mg/dL, >=100 mg/dL); Test type: Superiority; p < 0.001, Mixed Effect Model Repeat Measurement; LS-Mean Difference = 3.53, 95% CI 2-sided [3.02 to 4.03]

26. Secondary Outcome: Percent Change From Baseline in Log-Transformed Lipoprotein (a) (Lp[a]) and Triglycerides at Week 14
Time Frame: Baseline, Week 14
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 8390 | 8394
Percent Change
  Lp (a): number analyzed (Participants) | 5914 | 5916
  Lp (a) | -1.3 (28.81) | -33.9 (29.62)
  Triglycerides: number analyzed (Participants) | 6443 | 6433
  Triglycerides | 0.6 (32.84) | -18.9 (28.44)
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); Lp (a): LS- mean differences and associated 95% CI, and p-values were from an MMRM model on the difference of log-transformed observations through Week 52 with fixed effects for treatment group, visit, treatment group*visit interaction, log-transformed baseline value, log-transformed baseline value*visit interaction, geographical region and LDL-C at pre-screening (<100 mg/dL, >=100 mg/dL); Test type: Superiority; p < 0.001, Mixed Effect Model Repeat Measurement; LS-mean difference = 0.67, 95% CI 2-sided [0.66 to 0.68]
Statistical Analysis 2: Comparison: Placebo vs Bococizumab (PF-04950615); Triglycerides: LS- mean differences and associated 95% CI, and p-values were from an MMRM model through Week 70 on the difference of log-transformed observations with fixed effects for treatment group, visit, treatment group*visit interaction, log-transformed baseline value, log-transformed baseline value*visit interaction, geographical region and LDL-C at pre-screening (<100 mg/dL, >=100 mg/dL); Test type: Superiority; p < 0.001, Mixed Effect Model Repeat Measurement; LS-mean difference = 0.81, 95% CI 2-sided [0.80 to 0.81]

27. Secondary Outcome: Percent Change From Baseline in Log-Transformed High Sensitivity C-Reactive Protein (Hs-CRP) at Week 14
Time Frame: Baseline, Week 14
Population: Analysis was performed on FAS. Here, "N" signifies number of participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo | Bococizumab (PF-04950615)
Number analyzed (Participants) | 5931 | 5930
Percent change | -6.5 (88.28) | -1.1 (91.91)
Statistical Analysis 1: Comparison: Placebo vs Bococizumab (PF-04950615); LS- mean differences and associated 95% CI, and p-values were from an MMRM model on the difference of log-transformed observations through Week 52 with fixed effects for treatment group, visit, treatment group*visit interaction, log-transformed baseline value, log-transformed baseline value*visit interaction, geographical region and LDL-C at pre-screening (<100 mg/dL, >=100 mg/dL); Test type: Superiority; p < 0.001, Mixed Effect Model Repeat Measurement; LS-mean difference = 1.06, 95% CI 2-sided [1.03 to 1.10]

ADVERSE EVENTS:
Time Frame: Baseline up to 3.4 years
Description: Safety analysis set: all participants who randomized, had atleast 1 dose of study drug, excluding those attempted to randomize more than once in a bococizumab CV outcomes trial (B1481022/B1481038) or attempted to randomize in more than 1 CV outcomes trial, and all participants enrolled at study Site 3027 where a quality-related event was identified
Arm/Group | Placebo | Bococizumab (PF-04950615)
All-Cause Mortality (participants affected / at risk) | 65/8374 | 72/8386
Serious Adverse Events (participants affected / at risk) | 986/8374 | 1060/8386
Other Adverse Events (participants affected / at risk) | 1570/8374 | 2015/8386
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo (N=8374) | Bococizumab (PF-04950615) (N=8386)
Anaemia (Blood and lymphatic system disorders) | 8 | 6
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 2
Leukocytosis (Blood and lymphatic system disorders) | 2 | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 8 | 11
Acute left ventricular failure (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 29 | 40
Angina pectoris (Cardiac disorders) | 52 | 73
Angina unstable (Cardiac disorders) | 84 | 65
Aortic valve stenosis (Cardiac disorders) | 2 | 2
Arrhythmia (Cardiac disorders) | 1 | 3
Arteriosclerosis coronary artery (Cardiac disorders) | 4 | 2
Atrial fibrillation (Cardiac disorders) | 32 | 27
Atrial flutter (Cardiac disorders) | 9 | 3
Atrial tachycardia (Cardiac disorders) | 0 | 1
Atrial thrombosis (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 4
Atrioventricular block second degree (Cardiac disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 3 | 7
Cardiac arrest (Cardiac disorders) | 3 | 8
Cardiac discomfort (Cardiac disorders) | 1 | 0
Cardiac disorder (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 19 | 21
Cardiac failure acute (Cardiac disorders) | 2 | 3
Cardiac failure chronic (Cardiac disorders) | 1 | 2
Cardiac failure congestive (Cardiac disorders) | 32 | 24
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 4
Coronary artery disease (Cardiac disorders) | 31 | 30
Coronary artery dissection (Cardiac disorders) | 0 | 1
Coronary artery insufficiency (Cardiac disorders) | 0 | 1
Coronary artery occlusion (Cardiac disorders) | 5 | 1
Coronary artery stenosis (Cardiac disorders) | 4 | 5
Heart valve incompetence (Cardiac disorders) | 1 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 2 | 4
Left ventricular failure (Cardiac disorders) | 1 | 2
Microvascular coronary artery disease (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 32 | 35
Myocardial ischaemia (Cardiac disorders) | 6 | 6
Palpitations (Cardiac disorders) | 2 | 2
Pericardial effusion (Cardiac disorders) | 0 | 2
Pericarditis (Cardiac disorders) | 1 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 2
Sinus node dysfunction (Cardiac disorders) | 0 | 2
Sinus tachycardia (Cardiac disorders) | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 6
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 2
Ventricular arrhythmia (Cardiac disorders) | 0 | 2
Ventricular dysfunction (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 3
Ventricular tachycardia (Cardiac disorders) | 9 | 4
Hereditary haemorrhagic telangiectasia (Congenital, familial and genetic disorders) | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 2 | 0
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 4 | 3
Vestibular disorder (Ear and labyrinth disorders) | 0 | 1
Hyperparathyroidism (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Thyroid mass (Endocrine disorders) | 0 | 2
Angle closure glaucoma (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 2 | 1
Diabetic retinopathy (Eye disorders) | 1 | 1
Lens dislocation (Eye disorders) | 0 | 1
Macular fibrosis (Eye disorders) | 0 | 1
Optic ischaemic neuropathy (Eye disorders) | 0 | 1
Retinal artery occlusion (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 3 | 1
Retinal exudates (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal hernia obstructive (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 7 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0
Anal polyp (Gastrointestinal disorders) | 1 | 0
Anal prolapse (Gastrointestinal disorders) | 0 | 1
Appendix disorder (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Chronic gastritis (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 2 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 1
Colonic pseudo-obstruction (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 3
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Food poisoning (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 2 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 1
Gastric polyps (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 3
Gastritis erosive (Gastrointestinal disorders) | 1 | 1
Gastroduodenitis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 | 5
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal polyp haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 3
Gingival bleeding (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 2
Ileus (Gastrointestinal disorders) | 1 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 3
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 3 | 10
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Intestinal strangulation (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 3
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2
Mechanical ileus (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0
Necrotising colitis (Gastrointestinal disorders) | 0 | 1
Obstruction gastric (Gastrointestinal disorders) | 0 | 1
Oesophageal spasm (Gastrointestinal disorders) | 0 | 1
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 3
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 6 | 5
Peptic ulcer perforation (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 2
Rectal polyp (Gastrointestinal disorders) | 0 | 2
Salivary gland enlargement (Gastrointestinal disorders) | 0 | 1
Short-bowel syndrome (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Small intestinal stenosis (Gastrointestinal disorders) | 0 | 1
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 1 | 0
Tongue oedema (Gastrointestinal disorders) | 1 | 1
Ulcerative gastritis (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 1 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 3 | 0
Cardiac death (General disorders) | 1 | 0
Chest pain (General disorders) | 16 | 15
Death (General disorders) | 10 | 15
Electrocution (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 1
Generalised oedema (General disorders) | 0 | 1
Hyperplasia (General disorders) | 1 | 0
Ill-defined disorder (General disorders) | 1 | 0
Impaired healing (General disorders) | 1 | 0
Inflammation (General disorders) | 2 | 0
Injection site hypersensitivity (General disorders) | 0 | 1
Injection site reaction (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 3 | 3
Necrosis (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 47 | 45
Oedema peripheral (General disorders) | 0 | 1
Pain (General disorders) | 0 | 2
Pelvic mass (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 3
Sudden cardiac death (General disorders) | 1 | 3
Sudden death (General disorders) | 5 | 5
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Vascular stent restenosis (General disorders) | 1 | 4
Vascular stent thrombosis (General disorders) | 0 | 1
Bile duct stenosis (Hepatobiliary disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 2
Biliary colic (Hepatobiliary disorders) | 1 | 1
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 2
Cholecystitis (Hepatobiliary disorders) | 8 | 8
Cholecystitis acute (Hepatobiliary disorders) | 2 | 5
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 2
Cholecystocholangitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 3 | 8
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 1
Non-alcoholic fatty liver (Hepatobiliary disorders) | 0 | 1
Anaphylactic shock (Immune system disorders) | 1 | 1
Hypersensitivity (Immune system disorders) | 0 | 3
Abdominal abscess (Infections and infestations) | 1 | 0
Abdominal wall abscess (Infections and infestations) | 1 | 0
Abscess limb (Infections and infestations) | 0 | 2
Abscess neck (Infections and infestations) | 1 | 0
Acute sinusitis (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 3
Appendicitis (Infections and infestations) | 7 | 2
Arthritis bacterial (Infections and infestations) | 1 | 1
Arthritis infective (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 8 | 1
Bursitis infective (Infections and infestations) | 0 | 1
Bursitis infective staphylococcal (Infections and infestations) | 1 | 0
Carbuncle (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 13 | 11
Cellulitis of male external genital organ (Infections and infestations) | 0/6158 | 1/6180 — This is gender specific event.
Clostridium colitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 0
Creutzfeldt-Jakob disease (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Dermo-hypodermitis (Infections and infestations) | 1 | 0
Diabetic foot infection (Infections and infestations) | 1 | 4
Diverticulitis (Infections and infestations) | 7 | 5
Emphysematous pyelonephritis (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 2 | 1
Endocarditis bacterial (Infections and infestations) | 1 | 0
Endocarditis enterococcal (Infections and infestations) | 1 | 0
Endometritis (Infections and infestations) | 1 | 0
Epididymitis (Infections and infestations) | 2 | 0
Erysipelas (Infections and infestations) | 3 | 4
Furuncle (Infections and infestations) | 0 | 1
Gangrene (Infections and infestations) | 2 | 3
Gastritis viral (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 9 | 3
Gastroenteritis bacterial (Infections and infestations) | 1 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Groin abscess (Infections and infestations) | 1 | 1
H1N1 influenza (Infections and infestations) | 1 | 0
Haematoma infection (Infections and infestations) | 1 | 0
Hepatitis E (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 2 | 0
Incision site infection (Infections and infestations) | 1 | 0
Infected bite (Infections and infestations) | 2 | 0
Infected fistula (Infections and infestations) | 1 | 0
Infected seroma (Infections and infestations) | 2 | 0
Infected skin ulcer (Infections and infestations) | 1 | 1
Infectious pleural effusion (Infections and infestations) | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 3
Kidney infection (Infections and infestations) | 2 | 0
Klebsiella sepsis (Infections and infestations) | 0 | 1
Localised infection (Infections and infestations) | 1 | 3
Lower respiratory tract infection (Infections and infestations) | 2 | 2
Lower respiratory tract infection viral (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Lyme disease (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 8
Osteomyelitis bacterial (Infections and infestations) | 0 | 1
Osteomyelitis chronic (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 1 | 0
Penile infection (Infections and infestations) | 0 | 1
Periodontitis (Infections and infestations) | 0 | 1
Perirectal abscess (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 39 | 34
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pneumonia viral (Infections and infestations) | 2 | 0
Post procedural cellulitis (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0
Post procedural pneumonia (Infections and infestations) | 1 | 0
Prostatic abscess (Infections and infestations) | 1/6158 | 0/6180 — This is gender specific event.
Pyelonephritis (Infections and infestations) | 2 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 2
Pyomyositis (Infections and infestations) | 1 | 0
Rectal abscess (Infections and infestations) | 1 | 1
Respiratory tract infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 8 | 7
Sepsis syndrome (Infections and infestations) | 2 | 0
Septic shock (Infections and infestations) | 5 | 2
Skin candida (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 2
Streptococcal infection (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 2
Superinfection (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Tracheitis (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 3
Urinary tract infection (Infections and infestations) | 13 | 15
Urosepsis (Infections and infestations) | 5 | 3
Vestibular neuronitis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 1
Viral sepsis (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Visceral leishmaniasis (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 1 | 1
Wound infection staphylococcal (Infections and infestations) | 0 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 2
Arterial injury (Injury, poisoning and procedural complications) | 1 | 0
Brain herniation (Injury, poisoning and procedural complications) | 1 | 0
Burns second degree (Injury, poisoning and procedural complications) | 0 | 1
Cardiac function disturbance postoperative (Injury, poisoning and procedural complications) | 1 | 0
Cerebral ventricle collapse (Injury, poisoning and procedural complications) | 1 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 2 | 1
Concussion (Injury, poisoning and procedural complications) | 2 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 2
Coronary vascular graft occlusion (Injury, poisoning and procedural complications) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 2
Eye injury (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 6
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 3
Femur fracture (Injury, poisoning and procedural complications) | 0 | 4
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 2 | 1
Heat exhaustion (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 5 | 5
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 2
Incisional hernia (Injury, poisoning and procedural complications) | 2 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 1
Laceration (Injury, poisoning and procedural complications) | 0 | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 3 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 2
Mallet finger (Injury, poisoning and procedural complications) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 2
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 1
Patella fracture (Injury, poisoning and procedural complications) | 1 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 0 | 1
Post concussion syndrome (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 2
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Post procedural oedema (Injury, poisoning and procedural complications) | 1 | 0
Postoperative delirium (Injury, poisoning and procedural complications) | 0 | 1
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Procedural hypertension (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 2 | 0
Pubis fracture (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 4 | 4
Road traffic accident (Injury, poisoning and procedural complications) | 7 | 1
Seroma (Injury, poisoning and procedural complications) | 1 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 2
Soft tissue injury (Injury, poisoning and procedural complications) | 2 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 3
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 2 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 4 | 3
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 3 | 2
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 2 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 4 | 1
Vascular bypass dysfunction (Injury, poisoning and procedural complications) | 0 | 1
Vascular graft occlusion (Injury, poisoning and procedural complications) | 2 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 | 1
Vena cava injury (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 2
Alanine aminotransferase increased (Investigations) | 1 | 2
Aspartate aminotransferase increased (Investigations) | 1 | 2
Blood creatine phosphokinase increased (Investigations) | 1 | 2
Blood glucose decreased (Investigations) | 0 | 1
Blood glucose increased (Investigations) | 1 | 0
Blood pressure decreased (Investigations) | 0 | 1
Blood pressure diastolic decreased (Investigations) | 1 | 0
Cardiac stress test abnormal (Investigations) | 0 | 1
Electrocardiogram abnormal (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Heart rate abnormal (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Hepatitis C virus test positive (Investigations) | 0 | 1
International normalised ratio abnormal (Investigations) | 0 | 1
International normalised ratio decreased (Investigations) | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0
Liver function test increased (Investigations) | 0 | 5
Stress echocardiogram abnormal (Investigations) | 1 | 0
Weight decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 7
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 4
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 4 | 2
Diabetes with hyperosmolarity (Metabolism and nutrition disorders) | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 4 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 1
Hyperosmolar hyperglycaemic state (Metabolism and nutrition disorders) | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 5 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Insulin-requiring type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Obesity (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 4 | 4
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 6
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 5
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Diabetic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 6 | 4
Knee deformity (Musculoskeletal and connective tissue disorders) | 0 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 4
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3 | 10
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 18 | 22
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 3 | 6
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 2 | 3
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 2
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 2
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Anal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Benign gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 4
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Bladder transitional cell carcinoma stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cholesteatoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Colon cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intraocular melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Large cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lip and/or oral cavity cancer stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 5
Lung squamous cell carcinoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Maxillofacial sinus neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nasal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/2216 | 1/2206 — This is gender specific event.
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12/6158 | 13/6180 — This is gender specific event.
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/6158 | 1/6180 — This is gender specific event.
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/6158 | 0/6180 — This is gender specific event.
Rectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Renal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Soft tissue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of the cervix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/2216 | 0/2206 — This is gender specific event.
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/2216 | 1/2206 — This is gender specific event.
Axonal neuropathy (Nervous system disorders) | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Basal ganglia haemorrhage (Nervous system disorders) | 1 | 0
Brain stem infarction (Nervous system disorders) | 1 | 0
Carotid arteriosclerosis (Nervous system disorders) | 0 | 1
Carotid artery disease (Nervous system disorders) | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 8 | 14
Carpal tunnel syndrome (Nervous system disorders) | 0 | 2
Cauda equina syndrome (Nervous system disorders) | 1 | 1
Cerebellar haemorrhage (Nervous system disorders) | 1 | 1
Cerebellar infarction (Nervous system disorders) | 0 | 1
Cerebral artery occlusion (Nervous system disorders) | 2 | 0
Cerebral haematoma (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 2 | 3
Cerebral infarction (Nervous system disorders) | 1 | 3
Cerebral venous thrombosis (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 6 | 3
Cervical radiculopathy (Nervous system disorders) | 1 | 0
Chorea (Nervous system disorders) | 1 | 0
Coma (Nervous system disorders) | 1 | 0
Cubital tunnel syndrome (Nervous system disorders) | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 3 | 8
Embolic stroke (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 2 | 0
Epilepsy (Nervous system disorders) | 0 | 4
Facial paresis (Nervous system disorders) | 1 | 2
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Haemorrhagic cerebral infarction (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 2 | 2
Headache (Nervous system disorders) | 1 | 4
Hemiparesis (Nervous system disorders) | 1 | 3
Hypoaesthesia (Nervous system disorders) | 1 | 1
Hypoglycaemic coma (Nervous system disorders) | 1 | 0
Intraventricular haemorrhage (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 28 | 20
Lacunar infarction (Nervous system disorders) | 1 | 0
Lacunar stroke (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 3 | 0
Lumbar radiculopathy (Nervous system disorders) | 1 | 1
Lumbosacral radiculopathy (Nervous system disorders) | 0 | 2
Migraine (Nervous system disorders) | 0 | 1
Nerve compression (Nervous system disorders) | 3 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 1
Partial seizures (Nervous system disorders) | 1 | 1
Polyneuropathy (Nervous system disorders) | 0 | 1
Post stroke epilepsy (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 6 | 4
Radiculopathy (Nervous system disorders) | 2 | 0
Sciatica (Nervous system disorders) | 2 | 3
Seizure (Nervous system disorders) | 6 | 3
Syncope (Nervous system disorders) | 13 | 17
Thalamus haemorrhage (Nervous system disorders) | 1 | 0
Transient global amnesia (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 19 | 21
Vascular dementia (Nervous system disorders) | 1 | 0
Vertigo CNS origin (Nervous system disorders) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0/2216 | 1/2206 — This is gender specific event.
Device battery issue (Product Issues) | 0 | 1
Device dislocation (Product Issues) | 2 | 3
Acute psychosis (Psychiatric disorders) | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0
Alcoholism (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 2 | 1
Conversion disorder (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 2 | 0
Depression (Psychiatric disorders) | 2 | 4
Depression suicidal (Psychiatric disorders) | 0 | 1
Factitious disorder (Psychiatric disorders) | 0 | 1
Major depression (Psychiatric disorders) | 1 | 2
Mental status changes (Psychiatric disorders) | 1 | 1
Personality disorder (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 2
Suicide attempt (Psychiatric disorders) | 1 | 2
Acute kidney injury (Renal and urinary disorders) | 18 | 14
Acute prerenal failure (Renal and urinary disorders) | 1 | 0
Calculus urethral (Renal and urinary disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 2 | 2
Cystitis noninfective (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 2 | 3
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Ischaemic nephropathy (Renal and urinary disorders) | 0 | 1
Nephritis (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 4 | 6
Nephropathy (Renal and urinary disorders) | 1 | 0
Renal artery stenosis (Renal and urinary disorders) | 1 | 0
Renal cortical necrosis (Renal and urinary disorders) | 1 | 0
Renal disorder (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 3 | 2
Renal impairment (Renal and urinary disorders) | 2 | 0
Renal ischaemia (Renal and urinary disorders) | 1 | 0
Stag horn calculus (Renal and urinary disorders) | 0 | 1
Stress urinary incontinence (Renal and urinary disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 4 | 2
Urethral obstruction (Renal and urinary disorders) | 0 | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 2
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 5/6158 | 1/6180 — This is gender specific event.
Cystocele (Reproductive system and breast disorders) | 1/2216 | 0/2206 — This is gender specific event.
Fallopian tube obstruction (Reproductive system and breast disorders) | 0/2216 | 1/2206 — This is gender specific event.
Genital prolapse (Reproductive system and breast disorders) | 0/2216 | 1/2206 — This is gender specific event.
Menorrhagia (Reproductive system and breast disorders) | 1/2216 | 0/2206 — This is gender specific event.
Ovarian cyst (Reproductive system and breast disorders) | 1/2216 | 0/2206 — This is gender specific event.
Prostatic dysplasia (Reproductive system and breast disorders) | 1/6158 | 0/6180 — This is gender specific event.
Prostatic obstruction (Reproductive system and breast disorders) | 0/6158 | 1/6180 — This is gender specific event.
Prostatitis (Reproductive system and breast disorders) | 1/6158 | 1/6180 — This is gender specific event.
Prostatomegaly (Reproductive system and breast disorders) | 1/6158 | 0/6180 — This is gender specific event.
Rectocele (Reproductive system and breast disorders) | 1/2216 | 0/2206 — This is gender specific event.
Uterine polyp (Reproductive system and breast disorders) | 0/2216 | 1/2206 — This is gender specific event.
Uterine prolapse (Reproductive system and breast disorders) | 1/2216 | 0/2206 — This is gender specific event.
Vaginal haemorrhage (Reproductive system and breast disorders) | 1/2216 | 0/2206 — This is gender specific event.
Vaginal prolapse (Reproductive system and breast disorders) | 0/2216 | 1/2206 — This is gender specific event.
Vaginal ulceration (Reproductive system and breast disorders) | 0/2216 | 1/2206 — This is gender specific event.
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchial disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 11 | 22
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 10
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 8
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 2
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 2
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 2
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 4
Pregnancy of partner (Social circumstances) | 1/6158 | 1/6180 — This is gender specific event.
Hospitalisation (Surgical and medical procedures) | 0 | 1
Accelerated hypertension (Vascular disorders) | 1 | 0
Aneurysm (Vascular disorders) | 1 | 1
Aortic aneurysm (Vascular disorders) | 9 | 5
Aortic stenosis (Vascular disorders) | 1 | 1
Arterial stenosis (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 2 | 2
Arteriovenous fistula (Vascular disorders) | 0 | 1
Arteritis (Vascular disorders) | 1 | 1
Brachiocephalic vein stenosis (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 2 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 1
Dry gangrene (Vascular disorders) | 0 | 1
Embolism arterial (Vascular disorders) | 1 | 0
Extremity necrosis (Vascular disorders) | 1 | 0
Femoral artery aneurysm (Vascular disorders) | 0 | 1
Granulomatosis with polyangiitis (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 2 | 2
Hypertension (Vascular disorders) | 6 | 8
Hypertensive crisis (Vascular disorders) | 3 | 2
Hypertensive emergency (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 6 | 8
Hypovolaemic shock (Vascular disorders) | 0 | 1
Iliac artery occlusion (Vascular disorders) | 1 | 0
Infarction (Vascular disorders) | 1 | 0
Intermittent claudication (Vascular disorders) | 4 | 1
Ischaemia (Vascular disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 2 | 0
Orthostatic hypotension (Vascular disorders) | 2 | 2
Peripheral arterial occlusive disease (Vascular disorders) | 7 | 11
Peripheral artery aneurysm (Vascular disorders) | 0 | 1
Peripheral artery dissection (Vascular disorders) | 1 | 0
Peripheral artery occlusion (Vascular disorders) | 2 | 1
Peripheral artery stenosis (Vascular disorders) | 5 | 12
Peripheral ischaemia (Vascular disorders) | 4 | 9
Peripheral vascular disorder (Vascular disorders) | 7 | 8
Peripheral venous disease (Vascular disorders) | 1 | 0
Post thrombotic syndrome (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 0 | 1
Subclavian artery occlusion (Vascular disorders) | 1 | 0
Subclavian artery stenosis (Vascular disorders) | 1 | 0
Varicose vein (Vascular disorders) | 1 | 0
Vasculitis (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=8374) | Bococizumab (PF-04950615) (N=8386)
Diarrhoea (Gastrointestinal disorders) | 133 | 169
Injection site reaction (General disorders) | 88 | 588
Nasopharyngitis (Infections and infestations) | 289 | 283
Upper respiratory tract infection (Infections and infestations) | 193 | 183
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 195 | 217
Arthralgia (Musculoskeletal and connective tissue disorders) | 197 | 208
Back pain (Musculoskeletal and connective tissue disorders) | 203 | 217
Myalgia (Musculoskeletal and connective tissue disorders) | 160 | 170
Headache (Nervous system disorders) | 136 | 171
Hypertension (Vascular disorders) | 303 | 270

LIMITATIONS AND CAVEATS:
As specified in statistical analysis plan, due to discontinuation of the bococizumab clinical development program, health care resource utilization endpoints were not evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-02-12): https://cdn.clinicaltrials.gov/large-docs/76/NCT01975376/Prot_000.pdf
  • Statistical Analysis Plan (2016-12-20): https://cdn.clinicaltrials.gov/large-docs/76/NCT01975376/SAP_001.pdf